CLINICAL TRIAL: NCT01915498
Title: A Phase 1/2, Multicenter, Open-Label, Dose-Escalation and Expansion, Safety, Pharmacokinetic, Pharmacodynamic, and Clinical Activity Study of Orally Administered AG-221 in Subjects With Advanced Hematologic Malignancies With an IDH2 Mutation
Brief Title: Phase 1/2 Study of Enasidenib (AG-221) in Adults With Advanced Hematologic Malignancies With an Isocitrate Dehydrogenase Isoform 2 (IDH2) Mutation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Collaborators: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AG-221-C-001; 2013-001784-23 (EudraCT Number)
Record Dates: First submitted 2013-07-31; First posted 2013-08-05 (Estimated); Results first posted 2020-10-23 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-09

CONDITIONS: Hematologic Neoplasms
Keywords: acute myeloid leukemia; AML; myelodysplastic syndrome; MDS; hematologic malignancies; IDH2; Phase I; Phase II; AG-221; relapse AML; refractory AML
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — enasidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- enasidenib (Experimental): enasidenib administered orally. Multiple doses will be administered to determine the RP2D.
  Interventions: Drug: Enasidenib

INTERVENTIONS:
Drug: Enasidenib — Enasidenib tablets administered orally every day of 28-day treatment cycles until disease progression or unacceptable toxicities.
  Other Names: AG-221; IDHIFA

SUMMARY:
The primary objectives of Phase 1 Dose Escalation/Part 1 Expansion are:

* To assess the safety and tolerability of treatment with enasidenib administered continuously as a single agent dosed orally on Days 1 to 28 of a 28-day cycle in participants with advanced hematologic malignancies.
* To determine the maximum tolerated dose (MTD) or maximum administered dose (MAD) and/or the recommended Phase 2 dose (RP2D) of enasidenib in participants with advanced hematologic malignancies.

The primary objective of Phase 2 is:

• To assess the efficacy of enasidenib as treatment for participants with relapsed or refractory (R/R) acute myelogenous leukemia (AML) with an IDH2 mutation.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be greater than or equal to 18 years of age.
2. Subjects must have an advanced hematologic malignancy including:

Phase 1/ Dose escalation:

1. Diagnosis of acute myelogenous leukemia (AML) according to World Health Organization (WHO) criteria;

   * Disease refractory or relapsed (defined as the reappearance of > 5% blasts in the bone marrow).
   * Untreated AML, greater than or equal to 60 years of age and are not candidates for standard therapy due to age, performance status, and/or adverse risk factors, according to the treating physician and with approval of the Medical Monitor;
2. Diagnosis of Myelodysplastic syndrome (MDS) according to WHO classification with refractory anemia with excess blasts (RAEB-1 or RAEB-2), or considered high-risk by the Revised International Prognostic Scoring System (IPSS-R), that is recurrent or refractory, or the subject is intolerant to established therapy known to provide clinical benefit for their condition (i.e., subjects must not be candidates for regimens known to provide clinical benefit), according to the treating physician and with approval of the Medical Monitor.

   Phase 1/Part 1 Expansion:

   Arm 1: Relapsed or refractory AML and age greater than or equal to 60 years or any subject with AML regardless of age who has relapsed following a bone marrow transplant (BMT).

   Arm 2: Relapsed or refractory AML and age <60 years, excluding subjects with AML who have relapsed following a BMT.

   Arm 3: Untreated AML and age greater than or equal to 60 years that decline standard of care chemotherapy.

   Arm 4: Isocitrate dehydrogenase protein, 2 (IDH2)-mutated advanced hematologic malignancies not eligible for Arms 1 to 3.

   Phase 2:

   Diagnosis of AML according to World Health Organization (WHO) criteria and disease relapsed or refractory as defined by:
   * Subjects who relapse after allogeneic transplantation;
   * Subjects in second or later relapse;
   * Subjects who are refractory to initial induction or re-induction treatment
   * Subjects who relapse within 1 year of initial treatment, excluding patients with favorable-risk status according to National Comprehensive Cancer Network (NCCN) Guidelines. Favorable-risk cytogenetics: inv(16), t(16;16), t(8;21), t(15;17)
3. Subjects must have documented IDH2 gene-mutated disease:

   * For subjects in the dose escalation phase and Part 1 Expansion, IDH2 mutation may be based on local evaluation. (Centralized testing will be performed retrospectively.)
   * For subjects in the Phase 2 portion of the trial, central testing of IDH2 mutation of bone marrow aspirate and peripheral blood, is required during screening to confirm eligibility
4. Subjects must be amenable to serial bone marrow sampling, peripheral blood sampling and urine sampling during the study.

   * The diagnosis and evaluation of AML or MDS will be made by bone marrow aspiration and/or biopsy. If an aspirate is unobtainable (i.e., a "dry tap"), the diagnosis may be made from the core biopsy.
   * Screening bone marrow aspirate and peripheral blood samples are required of all subjects. A bone marrow biopsy must be collected if adequate aspirate is not attainable unless:

     * A bone marrow aspirate and biopsy was performed as part of the standard of care within 28 days prior to the start of the study treatment; and
     * Slides of bone marrow aspirate, biopsy and stained peripheral blood smear are available for both local and central pathology reviewers; and
     * A bone marrow aspirate sample acquired within 28 days prior to the start of study treatment has been sent for cytogenetic analysis.
5. Subjects must be able to understand and willing to sign an informed consent. A legally authorized representative may consent on behalf of a subject who is otherwise unable to provide informed consent, if acceptable to and approved by the site and/or sites Institutional Review Board (IRB)/Independent Ethics Committee (IEC).
6. Subjects must have Eastern Cooperative Oncology Group (ECOG) Performance status (PS) of 0 to 2.
7. Platelet count ≥ 20,000/μL (transfusions to achieve this level are allowed). Subjects with a baseline platelet count of < 20,000/μL due to underlying malignancy are eligible with Medical Monitor approval.
8. Subjects must have adequate hepatic function as evidenced by:

   * Serum total bilirubin ≤ 1.5 × upper limit of normal (ULN), unless considered due to Gilbert's disease, a gene mutation in UGT1A1, or leukemic organ involvement, following approval by the Medical Monitor;
   * Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase (ALP) ≤ 3.0 × ULN, unless considered due to leukemic organ involvement.
9. Subjects must have adequate renal function as evidenced by:

   • Serum creatinine ≤ 2.0 × ULN OR

   • Creatinine clearance greater than 40 mL/min based on the Cockroft-Gault glomerular filtration rate (GFR) estimation: (140 - Age) x (weight in kg) x (0.85 if female)/72 x serum creatinine
10. Subjects must be recovered from any clinically relevant toxic effects of any prior surgery, radiotherapy, or other therapy intended for the treatment of cancer. (Subjects with residual Grade 1 toxicity, for example Grade 1 peripheral neuropathy or residual alopecia, are allowed with approval of the Medical Monitor)
11. Female subjects of child-bearing potential must agree to undergo medically supervised pregnancy test prior to starting study drug. The first pregnancy test will be performed at screening (within 7 days prior to first study drug administration), and on the day of the first study drug administration and confirmed negative prior to dosing and Day 1 before dosing all subsequent cycles.
12. Female subjects with reproductive potential must have a negative serum pregnancy test within 7 days prior to the start of therapy. Subjects with reproductive potential are defined as sexually mature women who have not undergone a hysterectomy, bilateral oophorectomy or tubal occlusion or who have not been naturally postmenopausal (i.e., who have not menstruated at all) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months). Females of reproductive potential as well as fertile men and their partners who are female of reproductive potential must agree to abstain from sexual intercourse or to use two highly effective forms of contraception from the time of giving informed consent, during the study and for 120 days (females and males) following the last dose of AG-221. A highly effective form of contraception is defined as hormonal oral contraceptives, injectables, patches, intrauterine devices, double-barrier method (e.g., synthetic condoms, diaphragm, or cervical cap with spermicidal foam, cream, or gel), or male partner sterilization.
13. Able to adhere to the study visit schedule (ie, clinic visits at the study sites are mandatory, unless noted otherwise for particular study visits) and other protocol requirements.

Exclusion Criteria:

1. Subjects who have undergone hematopoietic stem cell transplant (HSCT) within 60 days of the first dose of AG-221, or subjects on immunosuppressive therapy post HSCT at the time of screening, or with clinically significant graft-versus-host disease (GVHD). (The use of a stable dose of oral steroids post GVHD and/or topical steroids for ongoing skin GVHD is permitted with Medical Monitor approval.)
2. Subjects who received systemic anticancer therapy or radiotherapy < 14 days prior to their first day of study drug administration. (Hydroxyurea is allowed for up to 28 days after the start of AG-221 for the control of peripheral leukemic blasts in subjects with white blood cell [WBC] counts > 30,000/μL as well as prior to enrollment).
3. Subjects who received a small molecule investigational agent < 14 days prior to their first day of study drug administration. In addition, the first dose of AG-221 should not occur before a period ≥ 5 half-lives of the investigational agent has elapsed.
4. Subjects taking the following sensitive cytochrome P450 (CYP) substrate medications that have a narrow therapeutic range are excluded from the study unless they can be transferred to other medications within ≥5 half-lives prior to dosing: paclitaxel (CYP2C8) warfarin, phenytoin (CYP2C9), S-mephenytoin (CYP2C19), thioridazine (CYP2D6), theophylline and tizanidine (CYP1A2).
5. Subjects taking the P-glycoprotein (P-gp) and breast cancer resistant protein (BCRP) transporter-sensitive substrates digoxin and rosuvastatin should be excluded from the study unless they can be transferred to other medications within ≥ 5 half-lives prior to dosing.
6. Subjects for whom potentially curative anticancer therapy is available.
7. Subjects who are pregnant or lactating.
8. Subjects with an active severe infection that required anti-infective therapy or with an unexplained fever > 38.5°C during screening visits or on their first day of study drug administration (at the discretion of the Investigator, subjects with tumor fever may be enrolled).
9. Subjects with known hypersensitivity to any of the components of AG-221.
10. Subjects with New York Heart Association (NYHA) Class III or IV congestive heart failure or left ventricular ejection fraction (LVEF) < 40% by echocardiogram (ECHO) or multi-gated acquisition (MUGA) scan within approximately 28 days of Cycle 1, Day 1 (C1D1).
11. Subjects with a history of myocardial infarction within the last 6 months of screening.
12. Subjects with uncontrolled hypertension (systolic blood pressure [BP] >180 mmHg or diastolic BP > 100 mmHg) at screening are excluded. Subjects requiring 2 or more medications to control hypertension are eligible with Medical Monitor approval.
13. Subjects with known unstable or uncontrolled angina pectoris.
14. Subjects with a known history of severe and/or uncontrolled ventricular arrhythmias.
15. Subjects with heart-rate corrected QT (QTc) interval ≥ 450 msec or other factors that increase the risk of QT prolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome) at screening.
16. Subjects taking medications that are known to prolong the QT interval unless they can be transferred to other medications within ≥ 5 half-lives prior to dosing.
17. Subjects with known infection with human immunodeficiency virus (HIV) or active hepatitis B or C.
18. Subjects with any other medical or psychological condition, deemed by the Investigator to be likely to interfere with a subject's ability to sign informed consent, cooperate, or participate in the study.
19. Subjects with known dysphagia, short-gut syndrome, gastroparesis, or other conditions that limit the ingestion or gastrointestinal absorption of drugs administered orally.
20. Subjects with clinical symptoms suggesting active central nervous system (CNS) leukemia or known CNS leukemia.
21. Subjects with immediately life-threatening, severe complications of leukemia such as uncontrolled bleeding, pneumonia with hypoxia or shock, and/or disseminated intravascular coagulation.
22. In the Phase 2 portion of the trial only, subjects who have previously received treatment with an inhibitor of Isocitrate dehydrogenase ( IDH).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2013-08-27 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (24):
- United States (19):
  - City Of Hope, Duarte, California
  - Stanford Cancer Center, Stanford, California
  - University Of Colorado Cancer Center, Aurora, Colorado
  - University of Miami Sylvester Cancer Center, Miami, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber/Mass General Brigham Cancer Care, Inc, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Cornell University Weill Medical College, New York, New York
  - Memorial Sloan-Kettering Cancer Center - NYC, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Gahanna, Ohio
  - Oregon Health and Science University OHSU, Portland, Oregon
  - Sarah Cannon Research Institute Drug Development Unit, Nashville, Tennessee
  - Ut Southwestern Medical Center At Dallas, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
- France (5):
  - Local Institution - 202, Bordeaux
  - Local Institution - 204, Paris
  - Local Institution - 203, Pessac
  - Local Institution - 205, Toulouse
  - Local Institution - 201, Villejuif

REFERENCES:
- [Background] Stein EM, DiNardo CD, Pollyea DA, Fathi AT, Roboz GJ, Altman JK, Stone RM, DeAngelo DJ, Levine RL, Flinn IW, Kantarjian HM, Collins R, Patel MR, Frankel AE, Stein A, Sekeres MA, Swords RT, Medeiros BC, Willekens C, Vyas P, Tosolini A, Xu Q, Knight RD, Yen KE, Agresta S, de Botton S, Tallman MS. Enasidenib in mutant IDH2 relapsed or refractory acute myeloid leukemia. Blood. 2017 Aug 10;130(6):722-731. doi: 10.1182/blood-2017-04-779405. Epub 2017 Jun 6. PMID 28588020
- [Background] Fathi AT, DiNardo CD, Kline I, Kenvin L, Gupta I, Attar EC, Stein EM, de Botton S; AG221-C-001 Study Investigators. Differentiation Syndrome Associated With Enasidenib, a Selective Inhibitor of Mutant Isocitrate Dehydrogenase 2: Analysis of a Phase 1/2 Study. JAMA Oncol. 2018 Aug 1;4(8):1106-1110. doi: 10.1001/jamaoncol.2017.4695. PMID 29346478
- [Background] Stein EM, DiNardo CD, Fathi AT, Pollyea DA, Stone RM, Altman JK, Roboz GJ, Patel MR, Collins R, Flinn IW, Sekeres MA, Stein AS, Kantarjian HM, Levine RL, Vyas P, MacBeth KJ, Tosolini A, VanOostendorp J, Xu Q, Gupta I, Lila T, Risueno A, Yen KE, Wu B, Attar EC, Tallman MS, de Botton S. Molecular remission and response patterns in patients with mutant-IDH2 acute myeloid leukemia treated with enasidenib. Blood. 2019 Feb 14;133(7):676-687. doi: 10.1182/blood-2018-08-869008. Epub 2018 Dec 3. PMID 30510081
- [Background] Pollyea DA, Tallman MS, de Botton S, Kantarjian HM, Collins R, Stein AS, Frattini MG, Xu Q, Tosolini A, See WL, MacBeth KJ, Agresta SV, Attar EC, DiNardo CD, Stein EM. Enasidenib, an inhibitor of mutant IDH2 proteins, induces durable remissions in older patients with newly diagnosed acute myeloid leukemia. Leukemia. 2019 Nov;33(11):2575-2584. doi: 10.1038/s41375-019-0472-2. Epub 2019 Apr 9. PMID 30967620
- [Background] Quek L, David MD, Kennedy A, Metzner M, Amatangelo M, Shih A, Stoilova B, Quivoron C, Heiblig M, Willekens C, Saada V, Alsafadi S, Vijayabaskar MS, Peniket A, Bernard OA, Agresta S, Yen K, MacBeth K, Stein E, Vassiliou GS, Levine R, De Botton S, Thakurta A, Penard-Lacronique V, Vyas P. Clonal heterogeneity of acute myeloid leukemia treated with the IDH2 inhibitor enasidenib. Nat Med. 2018 Aug;24(8):1167-1177. doi: 10.1038/s41591-018-0115-6. Epub 2018 Jul 16. PMID 30013198
- [Background] Amatangelo MD, Quek L, Shih A, Stein EM, Roshal M, David MD, Marteyn B, Farnoud NR, de Botton S, Bernard OA, Wu B, Yen KE, Tallman MS, Papaemmanuil E, Penard-Lacronique V, Thakurta A, Vyas P, Levine RL. Enasidenib induces acute myeloid leukemia cell differentiation to promote clinical response. Blood. 2017 Aug 10;130(6):732-741. doi: 10.1182/blood-2017-04-779447. Epub 2017 Jun 6. PMID 28588019
- [Background] Shih AH, Meydan C, Shank K, Garrett-Bakelman FE, Ward PS, Intlekofer AM, Nazir A, Stein EM, Knapp K, Glass J, Travins J, Straley K, Gliser C, Mason CE, Yen K, Thompson CB, Melnick A, Levine RL. Combination Targeted Therapy to Disrupt Aberrant Oncogenic Signaling and Reverse Epigenetic Dysfunction in IDH2- and TET2-Mutant Acute Myeloid Leukemia. Cancer Discov. 2017 May;7(5):494-505. doi: 10.1158/2159-8290.CD-16-1049. Epub 2017 Feb 13. PMID 28193779
- [Result] Stein EM, Fathi AT, DiNardo CD, Pollyea DA, Roboz GJ, Collins R, Sekeres MA, Stone RM, Attar EC, Frattini MG, Tosolini A, Xu Q, See WL, MacBeth KJ, de Botton S, Tallman MS, Kantarjian HM. Enasidenib in patients with mutant IDH2 myelodysplastic syndromes: a phase 1 subgroup analysis of the multicentre, AG221-C-001 trial. Lancet Haematol. 2020 Apr;7(4):e309-e319. doi: 10.1016/S2352-3026(19)30284-4. Epub 2020 Mar 5. PMID 32145771
- [Result] Intlekofer AM, Shih AH, Wang B, Nazir A, Rustenburg AS, Albanese SK, Patel M, Famulare C, Correa FM, Takemoto N, Durani V, Liu H, Taylor J, Farnoud N, Papaemmanuil E, Cross JR, Tallman MS, Arcila ME, Roshal M, Petsko GA, Wu B, Choe S, Konteatis ZD, Biller SA, Chodera JD, Thompson CB, Levine RL, Stein EM. Acquired resistance to IDH inhibition through trans or cis dimer-interface mutations. Nature. 2018 Jul;559(7712):125-129. doi: 10.1038/s41586-018-0251-7. Epub 2018 Jun 27. PMID 29950729
- [Result] Stein EM. Enasidenib, a targeted inhibitor of mutant IDH2 proteins for treatment of relapsed or refractory acute myeloid leukemia. Future Oncol. 2018 Jan;14(1):23-40. doi: 10.2217/fon-2017-0392. Epub 2017 Sep 18. PMID 29243965
- [Derived] Montesinos P, Fathi AT, de Botton S, Stein EM, Zeidan AM, Zhu Y, Prebet T, Vigil CE, Bluemmert I, Yu X, DiNardo CD. Differentiation syndrome associated with treatment with IDH2 inhibitor enasidenib: pooled analysis from clinical trials. Blood Adv. 2024 May 28;8(10):2509-2519. doi: 10.1182/bloodadvances.2023011914. PMID 38507688
- [Derived] de Botton S, Brandwein JM, Wei AH, Pigneux A, Quesnel B, Thomas X, Legrand O, Recher C, Chantepie S, Hunault-Berger M, Boissel N, Nehme SA, Frattini MG, Tosolini A, Marion-Gallois R, Wang JJ, Cameron C, Siddiqui M, Hutton B, Milkovich G, Stein EM. Improved survival with enasidenib versus standard of care in relapsed/refractory acute myeloid leukemia associated with IDH2 mutations using historical data and propensity score matching analysis. Cancer Med. 2021 Sep;10(18):6336-6343. doi: 10.1002/cam4.4182. Epub 2021 Aug 24. PMID 34427990
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/us/en/home.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 Dose Escalation: Enasidenib 30 mg BID: Participants received enasidenib 30 mg tablets twice a day (BID) on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Phase 1 Dose Escalation: Enasidenib 50 mg BID: Participants received enasidenib 50 mg tablets BID on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Phase 1 Dose Escalation: Enasidenib 75 mg BID: Participants received enasidenib 75 mg tablets BID on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Phase 1 Dose Escalation: Enasidenib 100 mg BID: Participants received enasidenib 100 mg tablets BID on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Phase 1 Dose Escalation: Enasidenib 150 mg BID: Participants received enasidenib 150 mg tablets BID on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Phase 1 Dose Escalation: Enasidenib 50 mg QD: Participants received enasidenib 50 mg tablets once a day (QD) on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Phase 1 Dose Escalation: Enasidenib 75 mg QD: Participants received enasidenib 75 mg tablets QD on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Phase 1 Dose Escalation: Enasidenib 100 mg QD: Participants received enasidenib 100 mg tablets QD on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Phase 1 Dose Escalation: Enasidenib 150 mg QD: Participants received enasidenib 150 mg tablets QD on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Phase 1 Dose Escalation: Enasidenib 200 mg QD: Participants received enasidenib 200 mg tablets QD on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Phase 1 Dose Escalation: Enasidenib 300 mg QD: Participants received enasidenib 300 mg tablets QD on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Phase 1 Dose Escalation: Enasidenib 450 mg QD: Participants received enasidenib 450 mg tablets QD on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Phase 1 Dose Escalation: Enasidenib 650 mg QD: Participants received enasidenib 650 mg tablets QD on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Phase 1 Dose Expansion Arm 1: Enasidenib 100 mg QD: Participants ≥ 60 years old with relapsed, refractory (R/R) AML or participants of any age if relapsed post-bone marrow transplant (BMT) received 100 mg enasidenib QD on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Phase 1 Dose Expansion Arm 2: Enasidenib 100 mg QD: Participants < 60 years old with R/R AML, excluding participants who relapsed post-BMT, received 100 mg enasidenib QD on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Phase 1 Dose Expansion Arm 3: Enasidenib 100 mg QD: Untreated AML participants ≥ 60 years old who declined standard of care received 100 mg enasidenib QD on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Phase 1 Dose Expansion Arm 4: Enasidenib 100 mg QD: Participants with advanced hematologic malignancies not eligible for Arms 1 to 3 received 100 mg enasidenib QD on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Phase 2: Enasidenib 100 mg QD: Participants received enasidenib 100 mg QD on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Safety Follow-Up: Enasidenib: Participants remaining on treatment as of the 01 September 2017 data cut-off date continued to receive enasidenib on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
Period: Main Analysis (Sept 2013 - Sept 2017)
Arm/Group | Phase 1 Dose Escalation: Enasidenib 30 mg BID | Phase 1 Dose Escalation: Enasidenib 50 mg BID | Phase 1 Dose Escalation: Enasidenib 75 mg BID | Phase 1 Dose Escalation: Enasidenib 100 mg BID | Phase 1 Dose Escalation: Enasidenib 150 mg BID | Phase 1 Dose Escalation: Enasidenib 50 mg QD | Phase 1 Dose Escalation: Enasidenib 75 mg QD | Phase 1 Dose Escalation: Enasidenib 100 mg QD | Phase 1 Dose Escalation: Enasidenib 150 mg QD | Phase 1 Dose Escalation: Enasidenib 200 mg QD | Phase 1 Dose Escalation: Enasidenib 300 mg QD | Phase 1 Dose Escalation: Enasidenib 450 mg QD | Phase 1 Dose Escalation: Enasidenib 650 mg QD | Phase 1 Dose Expansion Arm 1: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 2: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 3: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 4: Enasidenib 100 mg QD | Phase 2: Enasidenib 100 mg QD | Safety Follow-Up: Enasidenib
Started | 7 | 7 | 7 | 8 | 5 | 9 | 7 | 22 | 6 | 14 | 9 | 5 | 7 | 49 | 25 | 25 | 27 | 106 | 0
Completed (Completed indicates participants continuing treatment as of 01 September) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 2 | 3 | 6 | 0
Not Completed | 7 | 7 | 7 | 8 | 5 | 9 | 7 | 21 | 6 | 14 | 9 | 4 | 7 | 46 | 25 | 23 | 24 | 100 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 5 | 1 | 2 | 2 | 5 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 2 | 0
Not completed — Medical Condition | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Not completed — Development of Intercurrent Condition | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Not completed — Bone Marrow Transplant (BMT) | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 6 | 5 | 2 | 2 | 9 | 0
Not completed — Miscellaneous | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 4 | 8 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 2 | 1 | 1 | 1 | 1 | 2 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 4 | 1 | 4 | 3 | 16 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 4 | 1 | 2 | 1 | 1 | 2 | 4 | 1 | 4 | 2 | 16 | 0
Not completed — Disease Progression | 1 | 3 | 3 | 4 | 2 | 5 | 5 | 15 | 4 | 7 | 3 | 2 | 3 | 24 | 14 | 9 | 8 | 41 | 0
Period: Safety Follow-up (Sep 2017 to July 2019)
Arm/Group | Phase 1 Dose Escalation: Enasidenib 30 mg BID | Phase 1 Dose Escalation: Enasidenib 50 mg BID | Phase 1 Dose Escalation: Enasidenib 75 mg BID | Phase 1 Dose Escalation: Enasidenib 100 mg BID | Phase 1 Dose Escalation: Enasidenib 150 mg BID | Phase 1 Dose Escalation: Enasidenib 50 mg QD | Phase 1 Dose Escalation: Enasidenib 75 mg QD | Phase 1 Dose Escalation: Enasidenib 100 mg QD | Phase 1 Dose Escalation: Enasidenib 150 mg QD | Phase 1 Dose Escalation: Enasidenib 200 mg QD | Phase 1 Dose Escalation: Enasidenib 300 mg QD | Phase 1 Dose Escalation: Enasidenib 450 mg QD | Phase 1 Dose Escalation: Enasidenib 650 mg QD | Phase 1 Dose Expansion Arm 1: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 2: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 3: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 4: Enasidenib 100 mg QD | Phase 2: Enasidenib 100 mg QD | Safety Follow-Up: Enasidenib
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Ongoing Treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Period: Safety Follow up (Aug 2019 to Sep 2023)
Arm/Group | Phase 1 Dose Escalation: Enasidenib 30 mg BID | Phase 1 Dose Escalation: Enasidenib 50 mg BID | Phase 1 Dose Escalation: Enasidenib 75 mg BID | Phase 1 Dose Escalation: Enasidenib 100 mg BID | Phase 1 Dose Escalation: Enasidenib 150 mg BID | Phase 1 Dose Escalation: Enasidenib 50 mg QD | Phase 1 Dose Escalation: Enasidenib 75 mg QD | Phase 1 Dose Escalation: Enasidenib 100 mg QD | Phase 1 Dose Escalation: Enasidenib 150 mg QD | Phase 1 Dose Escalation: Enasidenib 200 mg QD | Phase 1 Dose Escalation: Enasidenib 300 mg QD | Phase 1 Dose Escalation: Enasidenib 450 mg QD | Phase 1 Dose Escalation: Enasidenib 650 mg QD | Phase 1 Dose Expansion Arm 1: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 2: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 3: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 4: Enasidenib 100 mg QD | Phase 2: Enasidenib 100 mg QD | Safety Follow-Up: Enasidenib
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set includes all participants who received at least one dose of study treatment.
Groups:
- Phase 1 Dose Expansion Arm 1: Enasidenib 100 mg QD: Participants ≥ 60 years old with relapsed or refractory AML or participants of any age if relapsed post-bone marrow transplant (BMT) received 100 mg enasidenib QD on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Phase 1 Dose Expansion Arm 2: Enasidenib 100 mg QD: Participants < 60 years old with relapsed, refractory AML, excluding participants who relapsed post-BMT, received 100 mg enasidenib QD on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Phase 1 Dose Escalation: Enasidenib 30 mg BID | Phase 1 Dose Escalation: Enasidenib 50 mg BID | Phase 1 Dose Escalation: Enasidenib 75 mg BID | Phase 1 Dose Escalation: Enasidenib 100 mg BID | Phase 1 Dose Escalation: Enasidenib 150 mg BID | Phase 1 Dose Escalation: Enasidenib 50 mg QD | Phase 1 Dose Escalation: Enasidenib 75 mg QD | Phase 1 Dose Escalation: Enasidenib 100 mg QD | Phase 1 Dose Escalation: Enasidenib 150 mg QD | Phase 1 Dose Escalation: Enasidenib 200 mg QD | Phase 1 Dose Escalation: Enasidenib 300 mg QD | Phase 1 Dose Escalation: Enasidenib 450 mg QD | Phase 1 Dose Escalation: Enasidenib 650 mg QD | Phase 1 Dose Expansion Arm 1: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 2: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 3: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 4: Enasidenib 100 mg QD | Phase 2: Enasidenib 100 mg QD | Total
Number analyzed (Participants) | 7 | 7 | 7 | 8 | 5 | 9 | 7 | 22 | 6 | 14 | 9 | 5 | 7 | 49 | 25 | 25 | 27 | 106 | 345
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (6.37) | 61.3 (8.86) | 64.7 (8.38) | 67.6 (12.88) | 73.6 (7.23) | 71.8 (9.00) | 62.3 (13.77) | 63.9 (15.06) | 73.8 (2.48) | 67.5 (14.69) | 68.3 (6.20) | 70.0 (8.77) | 70.1 (5.34) | 70.5 (11.09) | 49.2 (8.12) | 76.4 (6.87) | 68.1 (13.96) | 66.5 (11.88) | 66.8 (12.49)
Age, Customized [Count of Participants; unit: Participants]
  < 65 Years Old | 3 | 5 | 3 | 2 | 1 | 2 | 2 | 10 | 0 | 6 | 2 | 1 | 1 | 11 | 25 | 1 | 4 | 35 | 114
  ≥ 65- < 75 Years Old | 4 | 2 | 4 | 3 | 2 | 4 | 5 | 5 | 4 | 3 | 5 | 3 | 5 | 22 | 0 | 8 | 13 | 45 | 137
  ≥ 75 Years Old | 0 | 0 | 0 | 3 | 2 | 3 | 0 | 7 | 2 | 5 | 2 | 1 | 1 | 16 | 0 | 16 | 10 | 26 | 94
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 4 | 4 | 4 | 4 | 0 | 11 | 3 | 3 | 1 | 1 | 1 | 27 | 12 | 9 | 10 | 42 | 144
  Male | 4 | 2 | 3 | 4 | 1 | 5 | 7 | 11 | 3 | 11 | 8 | 4 | 6 | 22 | 13 | 16 | 17 | 64 | 201
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 7 | 3 | 2 | 1 | 8 | 27
  Not Hispanic or Latino | 4 | 6 | 5 | 7 | 3 | 8 | 3 | 15 | 6 | 8 | 8 | 4 | 4 | 36 | 16 | 22 | 19 | 60 | 234
  Unknown or Not Reported | 3 | 1 | 1 | 1 | 2 | 0 | 3 | 5 | 0 | 6 | 1 | 1 | 2 | 6 | 6 | 1 | 7 | 38 | 84
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6 | 6 | 6 | 6 | 2 | 6 | 5 | 18 | 6 | 11 | 8 | 4 | 5 | 40 | 17 | 24 | 19 | 78 | 267
  Black | 1 | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 4 | 0 | 0 | 6 | 19
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  American Indian/Alaskan Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Other | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 4
  Not Provided | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 4 | 0 | 2 | 1 | 1 | 1 | 6 | 2 | 1 | 6 | 21 | 50
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG performance status is used to describe a patient's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability (walking, working, etc.). The scale ranges from 0 to 5: -0 = Fully active, no restrictions; -1 = Restricted activity but ambulatory, able to carry out work of a light nature; -2 = Ambulatory and capable of all self-care but unable to carry out work activities; -3 = Limited self-care, confined to bed or chair more than 50% of waking hours; -4 = Completely disabled, no self-care, confined to bed or chair; -5 = Dead
  Participants
    0 - Fully active | 1 | 1 | 2 | 4 | 2 | 0 | 2 | 7 | 1 | 2 | 2 | 3 | 1 | 10 | 5 | 6 | 6 | 24 | 79
    1 - Restricted but ambulatory | 4 | 6 | 5 | 4 | 2 | 5 | 4 | 11 | 4 | 9 | 4 | 1 | 5 | 28 | 18 | 13 | 16 | 65 | 204
    2 - Ambulatory but unable to work | 2 | 0 | 0 | 0 | 1 | 4 | 1 | 4 | 1 | 3 | 3 | 1 | 1 | 11 | 2 | 6 | 5 | 16 | 61
    3 - Limited self-care | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    4 - Completely Disabled | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Isocitrate dehydrogenase 2 (IDH2) Mutation Type [Count of Participants; unit: Participants] — Isocitrate dehydrogenase 2 (IDH2) gene mutations have been described in patients with acute myeloid leukemia (AML) and myelodysplastic syndromes (MDS). Mutations in IDH2 most commonly lead to alterations affecting arginine-172 (R172) or arginine-140 (R140) in IDH2.
  Participants
    R140 | 6 | 6 | 6 | 5 | 2 | 6 | 6 | 19 | 5 | 10 | 9 | 1 | 5 | 37 | 18 | 17 | 21 | 80 | 259
    R172 | 1 | 1 | 1 | 3 | 2 | 3 | 1 | 3 | 1 | 4 | 0 | 4 | 2 | 12 | 7 | 8 | 5 | 26 | 84
    Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Missing | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Uridine Diphosphate-Glucuronosyltransferase 1 Family, Polypeptide A1 (UGT1A1) Mutation Status [Count of Participants; unit: Participants] — The UGT1A1 gene produces a protein, called the bilirubin uridine diphosphate glucuronosyl transferase (bilirubin-UGT) enzyme, an enzyme that glucuronidates bilirubin, a substance produced when red blood cells are broken down. This enzyme converts the toxic form of bilirubin (unconjugated bilirubin) to its nontoxic form (conjugated bilirubin), making it able to be dissolved and removed from the body. Enasidenib is an inhibitor of UGT1A1. Screening for UGT1A1 mutation was added in Protocol Amendment 4 therefore data are not not available for participants enrolled prior to Amendment 4.
  Participants
    Heterozygous | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 20 | 27
    Homozygous | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 1 | 10 | 16
    Wild Type | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 20 | 22
    Not Applicable | 7 | 7 | 7 | 7 | 5 | 9 | 7 | 21 | 4 | 14 | 8 | 5 | 6 | 47 | 24 | 21 | 23 | 36 | 258
    Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 20 | 22
Cytogenetic Risk Status [Count of Participants; unit: Participants] — Cytogenetic risk classification according to the National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines in Oncology for Acute Myeloid Leukemia. Risk categories are based on analysis of cytogenetics (the study of chromosomes), including chromosomal deletions, duplications, or substitutions and analysis of molecular abnormalities such as specific mutations. Better risk indicates disease more likely to respond to initial treatment and less likely to relapse whereas poor-risk is characterized by poor response to induction chemotherapy and higher relapse rates.
  Participants
    Favorable-Risk | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Intermediate-Risk | 4 | 5 | 1 | 2 | 1 | 5 | 2 | 6 | 4 | 9 | 6 | 3 | 3 | 19 | 14 | 13 | 19 | 57 | 173
    Poor-Risk | 1 | 1 | 2 | 2 | 2 | 3 | 1 | 8 | 1 | 2 | 0 | 1 | 3 | 13 | 8 | 8 | 2 | 26 | 84
    Failure | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 6 | 9
    Missing | 2 | 1 | 3 | 4 | 2 | 1 | 4 | 8 | 1 | 3 | 3 | 1 | 1 | 15 | 3 | 4 | 6 | 17 | 79
Bone Marrow Blasts [Count of Participants; unit: Participants]
  < 20% Blasts | 1 | 4 | 1 | 3 | 1 | 0 | 2 | 6 | 2 | 4 | 3 | 0 | 2 | 11 | 6 | 2 | 16 | 22 | 86
  20% to < 30% Blasts | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 4 | 2 | 6 | 2 | 14 | 34
  30% to < 50% Blasts | 5 | 2 | 1 | 2 | 1 | 2 | 0 | 5 | 2 | 5 | 2 | 2 | 1 | 8 | 4 | 6 | 3 | 18 | 69
  ≥ 50% Blasts | 1 | 1 | 4 | 3 | 2 | 6 | 4 | 11 | 1 | 4 | 3 | 3 | 4 | 26 | 12 | 10 | 6 | 49 | 150
  Missing | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 6
Malignancy Type [Count of Participants; unit: Participants]
  Relapsed / Refractory Acute Myeloid Leukemia (AML) | 6 | 7 | 6 | 6 | 3 | 8 | 5 | 19 | 3 | 9 | 8 | 3 | 7 | 48 | 25 | 3 | 9 | 105 | 280
  Untreated AML | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 3 | 0 | 2 | 0 | 1 | 0 | 22 | 5 | 1 | 39
  Myelodysplastic Syndrome (MDS) | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 3 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 17
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 9
Hemoglobin [Median (Full Range); unit: g/L] — Population: Participants with available data.
  g/L
    number analyzed (Participants) | 7 | 7 | 7 | 8 | 5 | 9 | 7 | 22 | 6 | 14 | 9 | 5 | 7 | 49 | 25 | 25 | 27 | 105 | 344
    (all) | 82.0 [72.0 to 95.0] | 97.0 [82.0 to 138.0] | 86.0 [76.0 to 111.0] | 97.5 [75.0 to 109.0] | 91.0 [75.0 to 93.0] | 89.0 [77.0 to 102.0] | 92.0 [73.0 to 110.0] | 96.5 [78.0 to 124.0] | 94.0 [79.0 to 132.0] | 87.5 [76.0 to 125.0] | 93.0 [78.0 to 131.0] | 103.0 [70.0 to 121.0] | 95.0 [76.0 to 122.0] | 93.0 [69.0 to 125.0] | 93.0 [70.0 to 129.0] | 89.0 [70.0 to 111.0] | 92.0 [71.0 to 152.0] | 89.0 [70.0 to 156.0] | 90.0 [69.0 to 156.0]
Platelets [Median (Full Range); unit: 10^9 cells/L] — Population: Participants with available data
  10^9 cells/L
    number analyzed (Participants) | 7 | 7 | 7 | 8 | 5 | 9 | 7 | 22 | 6 | 14 | 9 | 5 | 7 | 49 | 25 | 25 | 27 | 105 | 344
    (all) | 43.0 [15.0 to 147.0] | 91.0 [13.0 to 158.0] | 102.0 [17.0 to 167.0] | 92.0 [14.0 to 507.0] | 44.0 [26.0 to 183.0] | 23.0 [12.0 to 287.0] | 52.0 [8.0 to 253.0] | 35.5 [5.0 to 194.0] | 48.0 [12.0 to 72.0] | 42.0 [9.0 to 282.0] | 63.0 [21.0 to 486.0] | 73.0 [29.0 to 170.0] | 45.9 [17.0 to 247.0] | 39.0 [1.0 to 197.0] | 37.0 [6.0 to 292.0] | 58.0 [12.0 to 529.0] | 57.0 [13.0 to 644.0] | 36.0 [2.0 to 1288.0] | 42.9 [1.0 to 1228.0]
Absolute Neutrophil Count (ANC) [Median (Full Range); unit: 10^9 cells/L] — Population: Participants with available data
  10^9 cells/L
    number analyzed (Participants) | 7 | 6 | 6 | 8 | 5 | 9 | 7 | 22 | 6 | 12 | 9 | 5 | 7 | 49 | 25 | 23 | 27 | 105 | 338
    (all) | 0.8 [0.0 to 12.6] | 1.1 [0.4 to 4.7] | 0.5 [0.0 to 15.5] | 0.3 [0.0 to 2.0] | 0.5 [0.0 to 2.1] | 0.2 [0.0 to 3.4] | 0.2 [0.0 to 1.4] | 0.5 [0.0 to 32.1] | 1.0 [0.1 to 2.5] | 0.4 [0.1 to 7.4] | 0.6 [0.1 to 11.0] | 0.1 [0.1 to 1.1] | 0.8 [0.1 to 3.4] | 0.4 [0.0 to 5.4] | 0.1 [0.0 to 4.4] | 0.4 [0.0 to 6.7] | 1.0 [0.1 to 11.7] | 0.3 [0.0 to 70.0] | 0.4 [0.0 to 70.0]
White Blood Cell Count [Median (Full Range); unit: 10^9 cells/L] — Population: Participants with available data
  10^9 cells/L
    number analyzed (Participants) | 7 | 7 | 7 | 8 | 5 | 9 | 7 | 22 | 6 | 14 | 9 | 5 | 7 | 49 | 25 | 25 | 27 | 105 | 344
    (all) | 2.0 [0.6 to 57.2] | 2.1 [0.3 to 31.3] | 2.0 [0.2 to 39.7] | 2.5 [0.4 to 12.1] | 1.9 [1.5 to 16.8] | 2.6 [0.5 to 20.2] | 2.1 [0.5 to 14.7] | 5.3 [0.6 to 88.2] | 3.3 [0.8 to 26.9] | 2.6 [0.5 to 34.5] | 2.4 [0.7 to 47.9] | 1.3 [0.7 to 17.0] | 3.6 [0.8 to 38.3] | 3.0 [0.2 to 64.5] | 3.1 [0.4 to 26.9] | 2.3 [0.3 to 25.7] | 2.7 [0.4 to 26.7] | 2.0 [0.2 to 93.8] | 2.4 [0.2 to 93.8]

OUTCOME MEASURES:

1. Primary Outcome: Phase 1 Dose Escalation: Number of Participants With Dose Limiting Toxicities (DLT)
Description: Toxicity severity was graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.03. A DLT was defined as: • Non-hematologic toxicities: CTCAE ≥ Grade 3 with the exception of ≥ Grade 3 blood bilirubin increases in participants with a uridine diphosphate- glucuronosyltransferase 1 family, polypeptide A1 (UGT1A1) mutation. In participants with a UGT1A1 mutation, blood bilirubin increases of > 5× upper limit of normal (ULN) were considered a DLT. • Hematologic toxicities: Prolonged myelosuppression, defined as persistence of ≥ Grade 3 neutropenia or thrombocytopenia (by NCI CTCAE v4.03), leukemia-specific criteria, i.e., marrow cellularity <5% on Day 28 or later from the start of study drug without evidence of leukemia) at least 42 days after the initiation of Cycle 1 therapy. Leukemia-specific grading was used for cytopenias (based on percentage decrease from Baseline: 50 to 75% = Grade 3, >75% = Grade 4)
Time Frame: From time of first dose up to the end of Cycle 1; 28 days
Population: All participants who took at least one dose of study drug in the dose escalation phase and either had a DLT during Cycle 1, regardless of the amount of study drug exposure, or had no DLT and completed at least 75% of their planned Cycle 1 doses, and were considered to have had enough safety data to conclude that a DLT did not occur during Cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose Escalation: Enasidenib 30 mg BID | Phase 1 Dose Escalation: Enasidenib 50 mg BID | Phase 1 Dose Escalation: Enasidenib 75 mg BID | Phase 1 Dose Escalation: Enasidenib 100 mg BID | Phase 1 Dose Escalation: Enasidenib 150 mg BID | Phase 1 Dose Escalation: Enasidenib 50 mg QD | Phase 1 Dose Escalation: Enasidenib 75 mg QD | Phase 1 Dose Escalation: Enasidenib 100 mg QD | Phase 1 Dose Escalation: Enasidenib 150 mg QD | Phase 1 Dose Escalation: Enasidenib 200 mg QD | Phase 1 Dose Escalation: Enasidenib 300 mg QD | Phase 1 Dose Escalation: Enasidenib 450 mg QD | Phase 1 Dose Escalation: Enasidenib 650 mg QD
Number analyzed (Participants) | 4 | 5 | 5 | 7 | 4 | 0 | 0 | 5 | 6 | 6 | 4 | 5 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

2. Primary Outcome: Phase 1 Dose Escalation: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: A TEAE is any adverse event that began or worsened on or after the start of investigational product (IP) through 28 days after the last dose. A treatment-related TEAE is a TEAE that is suspected (possibly or probably related) by the Investigator to be related to the IP. A serious AE is one that at any dose of IP or at any time during the observation period met the following criteria: • Resulted in death; • Was life threatening; • Requires inpatient hospitalization or prolongation of existing hospitalization; • Resulted in persistent or significant disability/incapacity; • Was a congenital anomaly/birth defect; • Was medically important. The intensity of each AE was graded from 1 to 5 according to the NCI CTCAE Version 4.03, and according to the following: Mild (Grade 1), Moderate (Grade 2), Severe (Grade 3), Life threatening (Grade 4), or Death (Grade 5).
Time Frame: From the first dose of investigational product (IP) up to 28 days after the last dose, up to the data cutoff date of 01 September 2017; median treatment duration in the dose escalation phase was 5.0 months (range 0.4 to 34.2 months).
Population: The safety analysis set includes all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose Escalation: Enasidenib 30 mg BID | Phase 1 Dose Escalation: Enasidenib 50 mg BID | Phase 1 Dose Escalation: Enasidenib 75 mg BID | Phase 1 Dose Escalation: Enasidenib 100 mg BID | Phase 1 Dose Escalation: Enasidenib 150 mg BID | Phase 1 Dose Escalation: Enasidenib 50 mg QD | Phase 1 Dose Escalation: Enasidenib 75 mg QD | Phase 1 Dose Escalation: Enasidenib 100 mg QD | Phase 1 Dose Escalation: Enasidenib 150 mg QD | Phase 1 Dose Escalation: Enasidenib 200 mg QD | Phase 1 Dose Escalation: Enasidenib 300 mg QD | Phase 1 Dose Escalation: Enasidenib 450 mg QD | Phase 1 Dose Escalation: Enasidenib 650 mg QD
Number analyzed (Participants) | 7 | 7 | 7 | 8 | 5 | 9 | 7 | 22 | 6 | 14 | 9 | 5 | 7
Participants
  Any treatment-emergent adverse event (TEAE) | 7 | 7 | 7 | 8 | 5 | 9 | 7 | 22 | 6 | 14 | 9 | 5 | 7
  TEAE Related to Investigational Product (IP) | 6 | 7 | 6 | 5 | 5 | 3 | 3 | 17 | 6 | 14 | 7 | 4 | 7
  Grade 3-4 TEAE | 7 | 5 | 6 | 8 | 4 | 9 | 6 | 21 | 5 | 14 | 8 | 5 | 7
  Grade 3-4 TEAE Related to IP | 4 | 2 | 3 | 3 | 1 | 3 | 1 | 10 | 3 | 9 | 5 | 4 | 4
  Grade 5 TEAE | 4 | 1 | 2 | 2 | 2 | 3 | 1 | 5 | 0 | 2 | 4 | 2 | 0
  Grade 5 TEAE Related to IP | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Serious TEAE | 6 | 6 | 6 | 7 | 3 | 9 | 5 | 19 | 4 | 11 | 7 | 5 | 6
  Serious TEAE Related to IP | 2 | 4 | 2 | 2 | 0 | 2 | 1 | 9 | 1 | 5 | 3 | 2 | 2
  TEAE Leading to Discontinuation (D/C) of IP | 3 | 0 | 1 | 1 | 0 | 0 | 1 | 5 | 1 | 4 | 3 | 2 | 2
  TEAE Related to IP Leading to D/C of IP | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1
  TEAE Leading to Reduction of IP | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 3 | 1 | 3 | 6
  TEAE Related to IP Leading to Reduction of IP | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 3 | 6
  TEAE Leading to Interruption of IP | 4 | 1 | 3 | 5 | 2 | 6 | 0 | 10 | 2 | 9 | 3 | 3 | 6
  TEAE Related to IP Leading to Interruption of IP | 2 | 0 | 2 | 3 | 1 | 1 | 0 | 7 | 2 | 7 | 2 | 2 | 6

3. Primary Outcome: Phase 1 Dose Expansion: Number of Participants With Treatment Emergent Adverse Events
Description: A TEAE is any adverse event that began or worsened on or after the start of investigational product (IP) through 28 days after the last dose. A treatment-related TEAE is a TEAE that is suspected (possibly or probably related) by the Investigator to be related to the IP. A serious AE is one that at any dose of IP or at any time during the observation period met the following criteria: • Resulted in death; • Was life threatening; • Required inpatient hospitalization or prolongation of existing hospitalization; • Resulted in persistent or significant disability/incapacity; • Was a congenital anomaly/birth defect; • Was medically important. The intensity of each AE was graded from 1 to 5 according to the NCI CTCAE Version 4.03, and according to the following: Mild (Grade 1), Moderate (Grade 2), Severe (Grade 3), Life threatening (Grade 4), or Death (Grade 5).
Time Frame: From the first dose of investigational product (IP) up to 28 days after the last dose of IP up to the data cutoff date of 01 September 2017; median treatment duration in Part 1 Expansion was 5.2 months (range 0.5 to 32.8 months).
Population: All participants in Phase 1 Expansion who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose Expansion Arm 1: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 2: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 3: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 4: Enasidenib 100 mg QD
Number analyzed (Participants) | 49 | 25 | 25 | 27
Participants
  Any Treatment-emergent Adverse Event (TEAE) | 49 | 24 | 25 | 27
  TEAE Related to Investigational Product (IP) | 43 | 18 | 22 | 23
  Grade 3-4 TEAE | 47 | 21 | 21 | 20
  Grade 3-4 TEAE Related to IP | 20 | 9 | 15 | 7
  Grade 5 TEAE | 8 | 2 | 8 | 6
  Grade 5 TEAE Related to IP | 0 | 0 | 1 | 0
  Serious TEAE | 41 | 19 | 20 | 17
  Serious TEAE Related to IP | 7 | 6 | 8 | 2
  TEAE Leading to Discontinuation (D/C) of IP | 6 | 2 | 8 | 4
  TEAE Related to IP Leading to D/C of IP | 2 | 0 | 2 | 1
  TEAE Leading to Reduction of IP | 1 | 0 | 0 | 3
  TEAE Related to IP Leading to Reduction of IP | 0 | 0 | 0 | 3
  TEAE Leading to IP Interruption | 24 | 10 | 16 | 9
  TEAE Related to IP Leading to Interruption of IP | 9 | 3 | 7 | 3

4. Primary Outcome: Phase 2 Dose Expansion: Investigator Assessed Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants achieving an overall response of complete response (CR), CR with incomplete neutrophil recovery (CRi), CR with incomplete platelet recovery (CRp), partial response (PR), or morphologic leukemia-free state (MLFS) based on the 2003 revised International Working Group (IWG) criteria for AML, assessed by the Investigator. CR: • Absolute neutrophil count (ANC) > 1.0 x10⁹/L • Platelet count > 100 x10⁹/L • Bone marrow (BM) blasts < 5% • Absence of blasts with Auer rods • Independence of red cell transfusions CRi: • All CR criteria except for residual neutropenia (ANC < 1.0 x 10⁹/L CRp: • All CR criteria except for residual thrombocytopenia (platelets < 100 x 10⁹/L) PR: • Meets hematologic criteria of CR • Decrease of BM blasts to 5-25% and decrease of pretreatment BM blast ≥ 50%. MLFS: • Bone marrow blasts < 5% • Absence of blasts with Auer rods • Absence of extramedullary disease • No hematologic recovery required
Time Frame: Response assessments were performed every 28 days through Month 12 and every 56 days thereafter until the end of treatment; median duration of treatment exposure in Phase 2 was 5.3 months (range 0.4 to 22.5 months).
Population: All participants In Phase 2 with R/R AML who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Enasidenib 100 mg QD
Number analyzed (Participants) | 105
percentage of participants | 37.1 [27.9 to 47.1]

5. Primary Outcome: Phase 2 Dose Expansion: Number of Participants With Treatment Emergent Adverse Events
Description: A TEAE is any adverse event that began or worsened on or after the start of investigational product (IP) through 28 days after the last dose. A treatment-related TEAE is a TEAE that is suspected (possibly or probably related) by the Investigator to be related to the IP. A serious AE is one that at any dose of IP or at any time during the observation period met the following criteria: - Resulted in death; - Was life threatening; - Required inpatient hospitalization or prolongation of existing hospitalization; - Resulted in persistent or significant disability/incapacity; - Was a congenital anomaly/birth defect; - Was medically important. The intensity of each AE was graded from 1 to 5 according to the NCI CTCAE Version 4.03, and according to the following: Mild (Grade 1), Moderate (Grade 2), Severe (Grade 3), Life threatening (Grade 4), or Death (Grade 5).
Time Frame: From the first dose of investigational product (IP) up to 28 days after the last dose, up to the data cutoff of date of 01 September 2017; median duration of treatment exposure in Phase 2 was 5.3 months (range 0.4 to 22.5 months).
Population: All participants In Phase 2 with R/R AML who received at least 1 dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Enasidenib 100 mg QD
Number analyzed (Participants) | 105
Participants
  Any Treatment-emergent Adverse Event (TEAE) | 105
  TEAE Related to Investigational Product (IP) | 88
  Grade 3-4 TEAE | 92
  Grade 3-4 TEAE Related to IP | 48
  Grade 5 TEAE | 30
  Grade 5 TEAE Related to IP | 1
  Serious TEAE | 85
  Serious TEAE Related to IP | 34
  TEAE Leading to Discontinuation (D/C) of IP | 22
  TEAE Related to IP Leading to D/C of IP | 5
  TEAE Leading to Reduction of IP | 9
  TEAE Related to IP Leading to Reduction of IP | 7
  TEAE Leading to Interruption of IP | 49
  TEAE Related to IP Leading to Interruption of IP | 23

6. Primary Outcome: Safety Follow-up: Number of Participants With Treatment Emergent Adverse Events
Description: as for outcome 5
Time Frame: From the primary analysis cut-off date of 01 September 2017 to the final analysis cut-off date of 29 July 2019, a maximum of 23 months.
Population: Participants who received at least 1 dose of study treatment during the Safety Follow-up Period.
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Follow-up: Enasidenib
Number analyzed (Participants) | 16
Participants
  Any treatment-emergent adverse event (TEAE) | 16
  TEAE Related to Investigational Product (IP) | 6
  Grade 3-4 TEAE | 13
  Grade 3-4 TEAE Related to IP | 3
  Grade 5 TEAE | 0
  Grade 5 TEAE Related to IP | 0
  Serious TEAE | 9
  Serious TEAE Related to IP | 1
  TEAE Leading to Discontinuation (D/C) of IP | 0
  TEAE Related to IP Leading to D/C of IP | 0
  TEAE Leading to Reduction of IP | 0
  TEAE Related to IP Leading to Reduction of IP | 0
  TEAE Leading to Interruption of IP | 4
  TEAE Related to IP Leading to Interruption of IP | 0

7. Secondary Outcome: Phase 1 Dose Escalation: Investigator Assessed Overall Response Rate (ORR) by Total Daily Dose
Description: ORR is defined as the percentage of participants achieving an overall response of CR, CRi, CRp, PR, marrow CR (mCR) (for MDS) and MLFS (for AML) based on the 2003 revised IWG criteria for AML and 2006 modified IWG criteria for MDS. CR: • ANC > 1.0 x10⁹/L • Platelet count > 100 x10⁹/L • Bone marrow (BM) blasts < 5% • Absence of blasts with Auer rods • Independence of red cell transfusions CRi: • All CR criteria except for residual neutropenia (ANC < 1.0 x 10⁹/L CRp: • All CR criteria except for residual thrombocytopenia (platelet counts < 100 x 10⁹/L) PR: • Meets hematologic criteria of CR • Decrease of BM blasts to 5-25% and decrease of pretreatment BM blast ≥ 50%. MLFS: • Bone marrow blasts < 5% • Absence of blasts with Auer rods • Absence of extramedullary disease • No hematologic recovery required mCR: • Bone marrow myeloblasts ≤ 5% and decreased by ≥ 50%
Time Frame: Response assessments were performed every 28 days through Month 12 and every 56 days thereafter until the end of treatment; median duration of treatment exposure in the dose escalation phase was 5.0 months (range 0.4 to 34.2 months).
Population: All participants who received at least one dose of study treatment in Phase 1 Dose Escalation. Participants were grouped according to assigned total daily dose.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase 1 Dose Escalation: Enasidenib 50 mg: Participants received enasidenib 50 mg on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Phase 1 Dose Escalation: Enasidenib 60 mg: Participants who received a total daily dose of enasidenib 60 mg on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Phase 1 Dose Escalation: Enasidenib 75 mg: Participants who received a total daily dose of enasidenib 75 mg on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Phase 1 Dose Escalation: Enasidenib 100 mg: Participants who received a total daily dose of enasidenib 100 mg on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Phase 1 Dose Escalation: Enasidenib 150 mg: Participants who received a total daily dose of enasidenib 150 mg on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Phase 1 Dose Escalation: Enasidenib 200 mg: Participants who received a total daily dose of enasidenib 200 mg on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Phase 1 Dose Escalation: Enasidenib 300 mg: Participants who received a total daily dose of enasidenib 300 mg on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Phase 1 Dose Escalation: Enasidenib 450 mg: Participants who received a total daily dose of enasidenib 450 mg on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Phase 1 Dose Escalation: Enasidenib 650 mg: Participants who received a total daily dose of enasidenib 650 mg on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
Arm/Group | Phase 1 Dose Escalation: Enasidenib 50 mg | Phase 1 Dose Escalation: Enasidenib 60 mg | Phase 1 Dose Escalation: Enasidenib 75 mg | Phase 1 Dose Escalation: Enasidenib 100 mg | Phase 1 Dose Escalation: Enasidenib 150 mg | Phase 1 Dose Escalation: Enasidenib 200 mg | Phase 1 Dose Escalation: Enasidenib 300 mg | Phase 1 Dose Escalation: Enasidenib 450 mg | Phase 1 Dose Escalation: Enasidenib 650 mg
Number analyzed (Participants) | 9 | 7 | 7 | 29 | 13 | 22 | 14 | 5 | 7
percentage of participants | 33.3 [7.5 to 70.1] | 42.9 [9.9 to 81.6] | 14.3 [0.4 to 57.9] | 44.8 [26.4 to 64.3] | 46.2 [19.2 to 74.9] | 50.0 [28.2 to 71.8] | 35.7 [12.8 to 64.9] | 60.0 [14.7 to 94.7] | 71.4 [29.0 to 96.3]

8. Secondary Outcome: Phase 1 Dose Expansion: Investigator Assessed Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants achieving an overall response of CR, CRi, CRp, PR, mCR (for MDS), or MLFS (for AML) based on the 2003 revised IWG criteria for AML and 2006 modified IWG criteria for MDS. CR: - ANC > 1.0 x10⁹/L - Platelet count > 100 x10⁹/L - Bone marrow (BM) blasts < 5% - Absence of blasts with Auer rods - Independence of red cell transfusions CRi: - All CR criteria except for residual neutropenia (ANC < 1.0 x 10⁹/L CRp: - All CR criteria except for residual thrombocytopenia (platelet counts < 100 x 10⁹/L) PR: - Meets hematologic criteria of CR - Decrease of BM blasts to 5-25% and decrease of pretreatment BM blast ≥ 50%. MLFS: - Bone marrow blasts < 5% - Absence of blasts with Auer rods - Absence of extramedullary disease - No hematologic recovery required mCR: - Bone marrow myeloblasts ≤ 5% and decreased by ≥ 50%
Time Frame: Response assessments were performed every 28 days through Month 12 and every 56 days thereafter until the end of treatment; median duration of treatment exposure in Phase 1 Dose Expansion was 5.2 months (range 0.5 to 32.8 months).
Population: All participants who received at least one dose of study treatment in Phase 1 Expansion.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase 1 Dose Expansion Arm 1: Enasidenib 100 mg QD: Participants ≥ 60 years old with relapsed, refractory AML or participants of any age if relapsed post-bone marrow transplant (BMT) received 100 mg enasidenib QD on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
Arm/Group | Phase 1 Dose Expansion Arm 1: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 2: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 3: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 4: Enasidenib 100 mg QD
Number analyzed (Participants) | 49 | 25 | 25 | 27
percentage of participants | 46.9 [32.5 to 61.7] | 20.0 [6.8 to 40.7] | 36.0 [18.0 to 57.5] | 44.4 [25.5 to 64.7]

9. Secondary Outcome: Combined Phase 1/2: Investigator Assessed Overall Response Rate in Participants With R/R AML
Description: For participants with R/R AML ORR is defined as the percentage of participants achieving an overall response of CR, CRi, CRp, PR, or MLFS based on the 2003 revised IWG criteria for AML. CR: - ANC > 1.0 x10⁹/L - Platelet count > 100 x10⁹/L - Bone marrow (BM) blasts < 5% - Absence of blasts with Auer rods - Independence of red cell transfusions CRi: - All CR criteria except for residual neutropenia (ANC < 1.0 x 10⁹/L CRp: - All CR criteria except for residual thrombocytopenia (platelet counts < 100 x 10⁹/L) PR: - Meets hematologic criteria of CR - Decrease of BM blasts to 5-25% and decrease of pretreatment BM blast ≥ 50%. MLFS: - Bone marrow blasts < 5% - Absence of blasts with Auer rods - Absence of extramedullary disease - No hematologic recovery required
Time Frame: Response assessments were performed every 28 days through Month 12 and every 56 days thereafter until the end of treatment; median duration of treatment exposure for Phase 1 and 2 R/R AML participants was 5.4 months (range 0.4 to 34.2 months).
Population: All participants in Phase 1 and 2 with R/R AML who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Enasidenib 100 mg QD: Participants in Phase 1 or 2 with relapsed or refractory (R/R) AML who received enasidenib 100 mg QD on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
Arm/Group | Enasidenib 100 mg QD
Number analyzed (Participants) | 214
percentage of participants | 38.8 [32.2 to 45.7]

10. Secondary Outcome: Phase 1 Dose Escalation: Complete Response Rate (CRR) by Total Daily Dose
Description: Complete response rate is defined as the percentage of participants achieving a complete response (CR) based on the 2003 revised IWG criteria for AML or the 2006 modified IWG criteria for MDS as assessed by the investigator. CR for AML: - Absolute neutrophil count (ANC) > 1.0 x10⁹/L - Platelet count > 100 x10⁹/L - Bone marrow (BM) blasts < 5% - Absence of blasts with Auer rods - Independence of red cell transfusions CR for MDS: - Bone marrow: ≤ 5% myeloblasts with normal maturation of all cell lines - Peripheral blood: -- Hemoglobin ≥ 11 g/dL -- Platelets ≥ 100 × 10⁹/L -- Neutrophils ≥ 1.0 × 10⁹/L -- Blasts = 0%
Time Frame: Response assessments were performed every 28 days through Month 12 and every 56 days thereafter until the end of treatment; median duration of treatment exposure in Phase 1 Dose Escalation was 5.0 months (range 0.4 to 34.2 months).
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase 1 Dose Escalation: Enasidenib 50 mg: Participants received enasidenib 50 mg tablets QD on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
Arm/Group | Phase 1 Dose Escalation: Enasidenib 50 mg | Phase 1 Dose Escalation: Enasidenib 60 mg | Phase 1 Dose Escalation: Enasidenib 75 mg | Phase 1 Dose Escalation: Enasidenib 100 mg | Phase 1 Dose Escalation: Enasidenib 150 mg | Phase 1 Dose Escalation: Enasidenib 200 mg | Phase 1 Dose Escalation: Enasidenib 300 mg | Phase 1 Dose Escalation: Enasidenib 450 mg | Phase 1 Dose Escalation: Enasidenib 650 mg
Number analyzed (Participants) | 9 | 7 | 7 | 29 | 13 | 22 | 14 | 5 | 7
percentage of participants | 22.2 [2.8 to 60.0] | 14.3 [0.4 to 57.9] | 0.0 [0.0 to 41.0] | 27.6 [12.7 to 47.2] | 15.4 [1.9 to 45.4] | 4.5 [0.1 to 22.8] | 21.4 [4.7 to 50.8] | 40.0 [5.3 to 85.3] | 28.6 [3.7 to 71.0]

11. Secondary Outcome: Phase 1 Dose Expansion: Complete Response Rate
Description: as for outcome 10
Time Frame: as for outcome 8
Population: All participants in Phase 1 Dose Expansion who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1 Dose Expansion Arm 1: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 2: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 3: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 4: Enasidenib 100 mg QD
Number analyzed (Participants) | 49 | 25 | 25 | 27
percentage of participants | 22.4 [11.8 to 36.6] | 0.0 [0.0 to 13.7] | 20.0 [6.8 to 40.7] | 22.2 [8.6 to 42.3]

12. Secondary Outcome: Phase 2 Dose Expansion: Complete Response Rate
Description: Complete response rate is defined as the percentage of participants achieving a complete response (CR) based on the 2003 revised IWG criteria for AML as assessed by the investigator. CR for AML: - Absolute neutrophil count (ANC) > 1.0 x10⁹/L - Platelet count > 100 x10⁹/L - Bone marrow (BM) blasts < 5% - Absence of blasts with Auer rods - Independence of red cell transfusions
Time Frame: as for outcome 4
Population: All participants In Phase 2 with R/R AML who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Enasidenib 100 mg QD
Number analyzed (Participants) | 105
percentage of participants | 20.0 [12.8 to 28.9]

13. Secondary Outcome: Phase 1 Dose Escalation: Rate of Complete Response and Complete Response With Incomplete Hematological Recovery (CR/CRi/CRp) by Total Daily Dose
Description: The percentage of participants achieving a complete response (CR), CR with incomplete neutrophil recovery (CRi), or a CR with incomplete platelet recovery (CRp), based on the 2003 revised IWG criteria for AML and 2006 modified IWG criteria for MDS per investigator review. CR: - ANC > 1.0 x10⁹/L - Platelet count > 100 x10⁹/L - Bone marrow (BM) blasts < 5% - Absence of blasts with Auer rods - Independence of red cell transfusions CRi: - All CR criteria except for residual neutropenia (ANC < 1.0 x 10⁹/L CRp: - All CR criteria except for residual thrombocytopenia (platelet counts < 100 x 10⁹/L)
Time Frame: Response assessments were performed every 28 days through Month 12 and every 56 days thereafter until the end of treatment; median duration of treatment exposure in the Phase 1 Dose Escalation was 5.0 months (range 0.4 to 34.2 months).
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1 Dose Escalation: Enasidenib 50 mg | Phase 1 Dose Escalation: Enasidenib 60 mg | Phase 1 Dose Escalation: Enasidenib 75 mg | Phase 1 Dose Escalation: Enasidenib 100 mg | Phase 1 Dose Escalation: Enasidenib 150 mg | Phase 1 Dose Escalation: Enasidenib 200 mg | Phase 1 Dose Escalation: Enasidenib 300 mg | Phase 1 Dose Escalation: Enasidenib 450 mg | Phase 1 Dose Escalation: Enasidenib 650 mg
Number analyzed (Participants) | 9 | 7 | 7 | 29 | 13 | 22 | 14 | 5 | 7
percentage of participants | 22.2 [2.8 to 60.0] | 14.3 [0.4 to 57.9] | 0.0 [0.0 to 41.0] | 31.0 [15.3 to 50.8] | 15.4 [1.9 to 45.4] | 18.2 [5.2 to 40.3] | 28.6 [8.4 to 58.1] | 40.0 [5.3 to 85.3] | 57.1 [18.4 to 90.1]

14. Secondary Outcome: Phase 1 Dose Expansion: Rate of Complete Response and Complete Responses With Incomplete Hematological Recovery (CR/CRi/CRp)
Description: The percentage of participants achieving a complete response (CR), CR with incomplete neutrophil recovery (CRi), or a CR with incomplete platelet recovery (CRp) based on the 2003 revised IWG criteria for AML or the 2006 modified IWG criteria for MDS, assessed by the investigator. CR: - ANC > 1.0 x10⁹/L - Platelet count > 100 x10⁹/L - Bone marrow (BM) blasts < 5% - Absence of blasts with Auer rods - Independence of red cell transfusions CRi: - All CR criteria except for residual neutropenia (ANC < 1.0 x 10⁹/L CRp: - All CR criteria except for residual thrombocytopenia (platelet counts < 100 x 10⁹/L)
Time Frame: as for outcome 8
Population: All participants who received at least one dose of study treatment in Phase 1 Dose Expansion.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase 1 Dose Expansion Arm 1: Enasidenib 100 mg: Participants ≥ 60 years old with relapsed, refractory AML or participants of any age if relapsed post-bone marrow transplant (BMT) received 100 mg enasidenib QD on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
Arm/Group | Phase 1 Dose Expansion Arm 1: Enasidenib 100 mg | Phase 1 Dose Expansion Arm 2: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 3: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 4: Enasidenib 100 mg QD
Number analyzed (Participants) | 49 | 25 | 25 | 27
percentage of participants | 28.6 [16.6 to 43.3] | 8.0 [1.0 to 26.0] | 24.0 [9.4 to 45.1] | 25.9 [11.1 to 46.3]

15. Secondary Outcome: Phase 2 Dose Expansion: Rate of Complete Response and Complete Responses With Incomplete Hematological Recovery (CR/CRi/CRp)
Description: The percentage of participants achieving a complete response (CR), CR with incomplete neutrophil recovery (CRi), or a CR with incomplete platelet recovery (CRp) based on the 2003 revised IWG criteria for AML, assessed by the Investigator. CR: - ANC > 1.0 x10⁹/L - Platelet count > 100 x10⁹/L - Bone marrow (BM) blasts < 5% - Absence of blasts with Auer rods - Independence of red cell transfusions CRi: - All CR criteria except for residual neutropenia (ANC < 1.0 x 10⁹/L CRp: - All CR criteria except for residual thrombocytopenia (platelet counts < 100 x 10⁹/L)
Time Frame: as for outcome 4
Population: All participants In Phase 2 with R/R AML who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Enasidenib 100 mg QD
Number analyzed (Participants) | 105
percentage of participants | 31.4 [22.7 to 41.2]

16. Secondary Outcome: Phase 1 Dose Expansion: Kaplan-Meier Estimate of Duration of Response (DOR)
Description: Among participants who had a response of CR, CRi, CRp, PR, mCR, or MLFS based on the 2003 revised IWG criteria for AML or the 2006 modified IWG criteria for MDS, assessed by the Investigator, duration of response was calculated from the date of the first occurrence of response to the date of documented disease relapse, progression, or death due to any cause, whichever occurred first. DOR was estimated using the Kaplan-Meier method. Participants without relapse, progressive disease, or death due to any cause were censored at the date of the last adequate response assessment.
Time Frame: From first dose of study treatment to the data cut-off date of 01 September 2017; overall median time on follow-up in Phase 1 Dose Expansion was 8.3 months (range 0.5 to 32.8 months).
Population: Participants who received at least one dose of study treatment in Phase 1 Dose Expansion with an objective response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1 Dose Expansion Arm 1: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 2: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 3: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 4: Enasidenib 100 mg QD
Number analyzed (Participants) | 23 | 5 | 9 | 12
months | 5.6 [1.9 to 18.5] | 3.9 [1.9 to 5.1] | NA [1.9 to NA] — Not estimable due to low number of events | 12.0 [0.4 to NA] — Not estimable due to low number of events

17. Secondary Outcome: Phase 2 Dose Expansion: Kaplan-Meier Estimate of Duration of Response
Description: For participants with an objective response based on the 2003 revised IWG criteria for AML assessed by the Investigator, duration of response was calculated from the date of the first occurrence of response to the date of documented disease relapse, progression, or death due to any cause, whichever occurred first. Participants without relapse, progressive disease or death were censored at the last response assessment date. Relapse (for participants who previously attained CR, Cri, CRp or MLFS): BM blasts ≥ 5%, reappearance of blasts in the blood or development of extramedullary disease. Disease progression (for participants who previously attained PR): development of new extramedullary disease, or For participants with 5% to 67% BM blasts at nadir: - a > 50% increase in BM blasts from nadir and that is ≥ 20%. For participants with ≥ 67% BM blasts at nadir: - a doubling of the nadir absolute peripheral blood (PB) blast count and the final absolute PB blast count > 10 x 10⁹/L.
Time Frame: From first dose of study treatment to the data cut-off date of 01 September 2017; median time on follow-up in Phase 2 was 5.8 months (range 0.4 to 22.5 months).
Population: Participants in Phase 2 with R/R AML who received at least one dose of study treatment and who had an objective response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Enasidenib 100 mg QD
Number analyzed (Participants) | 39
months | 5.6 [3.7 to 7.4]

18. Secondary Outcome: Phase 1 Dose Expansion: Kaplan-Meier Estimate of Overall Survival
Description: Overall survival is defined as the time from first dose to the date of death due to any cause. Participants still alive were censored at the last date known to be alive or at the data cut-off date, whichever was earlier.
Time Frame: as for outcome 16
Population: All participants in Phase 1 Dose Expansion who received at least one dose of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1 Dose Expansion Arm 1: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 2: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 3: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 4: Enasidenib 100 mg QD
Number analyzed (Participants) | 49 | 25 | 25 | 27
months | 8.8 [7.5 to 10.5] | 11.6 [6.5 to 15.4] | 10.6 [6.2 to 19.8] | 11.3 [3.6 to 19.1]

19. Secondary Outcome: Phase 2 Dose Expansion: Kaplan-Meier Estimate of Overall Survival
Description: as for outcome 18
Time Frame: as for outcome 17
Population: All participants In Phase 2 with R/R AML who received at least 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Enasidenib 100 mg QD
Number analyzed (Participants) | 105
months | 7.0 [4.9 to 8.8]

20. Secondary Outcome: Phase 1 Combined: Percentage of Participants Who Achieved 56-Day Red Blood Cell Transfusion Independence Post-baseline
Description: Participants who achieved 56-day post-baseline red blood cell (RBC) transfusion independence, i.e. with no RBC transfusions for at least 56 consecutive days during the treatment exposure period, reported by Baseline RBC transfusion dependence status. Participants with at least one transfusion during the Baseline period were considered transfusion dependent at Baseline, where the Baseline period is defined as 28 days before and 28 days after the first dose of treatment for Phase 1. Results are reported for all participants in Phase 1 combined and for the subset of participants with R/R AML.
Time Frame: Baseline to the end of treatment; overall median duration of treatment exposure in Phase 1 combined was 5.1 months (range 0.4, 34.2 months).
Population: The population included all participants who received at least one dose of study treatment in Phase 1 Dose Escalation and Dose Expansion. Results were analyzed and are reported for Phase 1 combined.
Measure: Number; unit: percentage of participants
Groups:
- Phase 1: Enasidenib - R/R AML: Participants in Phase 1 Dose Escalation and Phase 1 Dose Expansion with R/R AML who received any dose of enasidenib on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Phase 1: Enasidenib: Participants in Phase 1 Dose Escalation and Phase 1 Dose Expansion who received any dose of enasidenib on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
Arm/Group | Phase 1: Enasidenib - R/R AML | Phase 1: Enasidenib
Number analyzed (Participants) | 175 | 239
percentage of participants
  Baseline Transfusion Dependent: number analyzed (Participants) | 135 | 182
  Baseline Transfusion Dependent | 39.3 | 38.5
  Baseline Transfusion Independent: number analyzed (Participants) | 40 | 57
  Baseline Transfusion Independent | 80.0 | 71.9

21. Secondary Outcome: Phase 1 Combined: Percentage of Participants Who Achieved 56-Day Platelet Transfusion Independence Post-baseline
Description: Participants who achieved 56-day post-baseline platelet transfusion independence, i.e. with no platelet transfusions for at least 56 consecutive days during the treatment exposure period, reported by Baseline platelet transfusion dependence status. Participants with at least one transfusion during the Baseline period were considered transfusion dependent at Baseline, where the Baseline period is defined as 28 days before and 28 days after the first dose of treatment for Phase 1. Results are reported for all participants in Phase 1 combined and for the subset of participants with R/R AML.
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1: Enasidenib - R/R AML | Phase 1: Enasidenib
Number analyzed (Participants) | 175 | 239
percentage of participants
  Baseline Transfusion Dependent: number analyzed (Participants) | 106 | 136
  Baseline Transfusion Dependent | 38.7 | 33.1
  Baseline Transfusion Independent: number analyzed (Participants) | 69 | 103
  Baseline Transfusion Independent | 78.3 | 76.7

22. Secondary Outcome: Phase 2: Percentage of Participants Who Achieved 56-Day Red Blood Cell Transfusion Independence Post-baseline
Description: Participants who achieved 56-day post-baseline red blood cell (RBC) transfusion independence, i.e. with no RBC transfusions for at least 56 consecutive days during the treatment exposure period, reported by Baseline RBC transfusion dependence status. Participants with at least one transfusion during the Baseline period were considered transfusion dependent at Baseline, where the Baseline period is defined as 56 days before the first dose date for Phase 2.
Time Frame: Baseline to the end of treatment; median duration of treatment exposure in Phase 2 was 5.3 months (range 0.4 to 22.5 months).
Population: All participants In Phase 2 with R/R AML who received at least 1 dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2: Enasidenib 100 mg QD
Number analyzed (Participants) | 105
percentage of participants
  Baseline Transfusion Dependent: number analyzed (Participants) | 67
  Baseline Transfusion Dependent | 41.8
  Baseline Transfusion Independent: number analyzed (Participants) | 38
  Baseline Transfusion Independent | 57.9

23. Secondary Outcome: Phase 2: Percentage of Participants Who Achieved 56-Day Platelet Transfusion Independence Post-baseline
Description: Participants who achieved 56-day post-baseline platelet transfusion independence, i.e. with no platelet transfusions for at least 56 consecutive days during the treatment exposure period, reported by Baseline platelet transfusion dependence status. Participants with at least one transfusion during the Baseline period were considered transfusion dependent at Baseline, where the Baseline period is defined as 56 days before the first dose date for Phase 2.
Time Frame: as for outcome 22
Population: All participants In Phase 2 with R/R AML who received at least 1 dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2: Enasidenib 100 mg QD
Number analyzed (Participants) | 105
percentage of participants
  Baseline Transfusion Dependent: number analyzed (Participants) | 59
  Baseline Transfusion Dependent | 35.6
  Baseline Transfusion Independent: number analyzed (Participants) | 46
  Baseline Transfusion Independent | 69.6

24. Secondary Outcome: Phase 1 Dose Expansion: Kaplan-Meier Estimate of Event Free Survival (EFS)
Description: Event-free survival is defined as the interval from the date of the first dose to the date of documented relapse, progression, or death due to any cause, whichever occurs first. Participants without an EFS event were censored at the date of the last adequate response assessment.
Time Frame: as for outcome 16
Population: All participants in Phase 1 Dose Expansion who received at least one dose of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1 Dose Expansion Arm 1: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 2: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 3: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 4: Enasidenib 100 mg QD
Number analyzed (Participants) | 49 | 25 | 25 | 27
months | 4.0 [3.8 to 7.0] | 3.8 [2.6 to 8.8] | 9.2 [2.8 to NA] — Not estimable due to the low number of events | 3.8 [1.8 to 11.3]

25. Secondary Outcome: Phase 2 Dose Expansion: Kaplan-Meier Estimate of Event Free Survival
Description: Event-free survival is defined as the interval from the date of the first dose to the date of documented relapse, progression, or death due to any cause, whichever occurred first. Participants without an EFS event were censored at the date of the last adequate response assessment.
Time Frame: as for outcome 17
Population: All participants In Phase 2 with R/R AML who received at least 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Enasidenib 100 mg QD
Number analyzed (Participants) | 105
months | 4.7 [3.0 to 5.6]

26. Secondary Outcome: Phase 1 Dose Expansion: Kaplan-Meier Estimate of Duration of Complete Response (DOCR)
Description: Among participants who had a response of CR based on the 2003 revised IWG criteria for AML and 2006 modified IWG criteria for MDS assessed by the Investigator, duration of complete response was calculated from the date of the first occurrence of complete response to the date of documented disease relapse, progression or death, whichever occurred earlier. DOCR was estimated using the Kaplan-Meier method. Participants without relapse, progressive disease, or death due to any cause were censored at the date of the last adequate response assessment.
Time Frame: as for outcome 16
Population: Participants who received at least one dose of study treatment in Phase 1 Dose Expansion with a complete response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1 Dose Expansion Arm 1: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 2: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 3: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 4: Enasidenib 100 mg QD
Number analyzed (Participants) | 11 | 0 | 5 | 6
months | 11.6 [1.9 to NA] — Not estimable due to low number of events |  | NA [3.7 to NA] — Not estimable due to low number of events | 16.8 [2.6 to NA] — Not estimable due to low number of events

27. Secondary Outcome: Phase 2 Dose Expansion: Duration of Complete Response
Description: Among participants who had a response of CR based on the 2003 revised IWG criteria for AML assessed by the Investigator, duration of complete response was calculated from the date of the first occurrence of complete response to the date of documented disease relapse, progression or death, whichever occurred earlier. DOCR was estimated using the Kaplan-Meier method. Participants without relapse, progressive disease, or death due to any cause were censored at the date of the last adequate response assessment.
Time Frame: as for outcome 17
Population: Participants in Phase 2 with R/R AML who received at least one dose of study treatment and who had a complete response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Enasidenib 100 mg QD
Number analyzed (Participants) | 21
months | 4.6 [2.8 to 6.5]

28. Secondary Outcome: Phase 1 Dose Escalation: Time to First Response by Total Daily Dose
Description: Time to response is defined as the time from the date of first dose to the date of the first occurrence of response of CR, CRi, CRp, PR, mCR (for MDS) or MLFS (for AML) based on the 2003 revised IWG criteria for AML and 2006 modified IWG criteria for MDS as assessed by the Investigator.
Time Frame: as for outcome 10
Population: Participants who received at least one dose of study treatment in Phase 1 Dose Escalation who had an objective response. Participants were grouped according to assigned total daily dose.
Measure: Median (Full Range); unit: months
Groups:
- Phase 1 Dose Escalation: Enasidenib 60 mg: Participants received enasidenib 60 mg on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Phase 1 Dose Escalation: Enasidenib 75 mg: Participants received enasidenib 75 mg on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Phase 1 Dose Escalation: Enasidenib 100 mg: Participants received enasidenib 100 mg on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Phase 1 Dose Escalation: Enasidenib 150 mg: Participants received enasidenib 150 mg on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Phase 1 Dose Escalation: Enasidenib 200 mg: Participants received enasidenib 200 mg on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Phase 1 Dose Escalation: Enasidenib 300 mg: Participants received enasidenib 300 mg on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Phase 1 Dose Escalation: Enasidenib 450 mg: Participants received enasidenib 450 mg on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Phase 1 Dose Escalation: Enasidenib 650 mg: Participants received enasidenib 650 mg on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
Arm/Group | Phase 1 Dose Escalation: Enasidenib 50 mg | Phase 1 Dose Escalation: Enasidenib 60 mg | Phase 1 Dose Escalation: Enasidenib 75 mg | Phase 1 Dose Escalation: Enasidenib 100 mg | Phase 1 Dose Escalation: Enasidenib 150 mg | Phase 1 Dose Escalation: Enasidenib 200 mg | Phase 1 Dose Escalation: Enasidenib 300 mg | Phase 1 Dose Escalation: Enasidenib 450 mg | Phase 1 Dose Escalation: Enasidenib 650 mg
Number analyzed (Participants) | 3 | 3 | 1 | 13 | 6 | 11 | 5 | 3 | 5
months | 3.8 [1.0 to 4.2] | 1.9 [1.0 to 3.8] | 0.9 [0.9 to 0.9] | 1.8 [0.6 to 5.6] | 2.0 [0.6 to 8.6] | 1.9 [0.5 to 5.7] | 2.1 [1.0 to 3.7] | 2.8 [0.5 to 3.8] | 1.9 [0.5 to 3.8]

29. Secondary Outcome: Phase 1 Dose Expansion: Time to First Response
Description: as for outcome 28
Time Frame: as for outcome 8
Population: Participants who received at least one dose of study treatment in Phase 1 Dose Expansion who had an objective response.
Measure: Median (Full Range); unit: months
Arm/Group | Phase 1 Dose Expansion Arm 1: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 2: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 3: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 4: Enasidenib 100 mg QD
Number analyzed (Participants) | 23 | 5 | 9 | 12
months | 1.9 [0.5 to 9.4] | 3.7 [0.9 to 5.5] | 1.8 [1.0 to 3.8] | 1.4 [0.5 to 9.2]

30. Secondary Outcome: Phase 2 Dose Expansion: Time to First Response
Description: Time to response is defined as the time from the date of first dose to the date of the first occurrence of response of CR, CRi, CRp, PR, or MLFS based on the 2003 revised IWG criteria for AML as assessed by the Investigator.
Time Frame: as for outcome 4
Population: as for outcome 17
Measure: Median (Full Range); unit: months
Arm/Group | Phase 2: Enasidenib 100 mg QD
Number analyzed (Participants) | 39
months | 2.7 [0.9 to 7.5]

31. Secondary Outcome: Phase 1 Dose Escalation: Time to Best Response by Total Daily Dose
Description: Time to best response is defined as the time from the date of the first dose to the date of the first occurrence of best response according to the following hierarchical order: CR, CRi/CRp, PR, mCR (for MDS) / MLFS (for AML) based on the 2003 revised IWG criteria for AML and 2006 modified IWG criteria for MDS per investigator assessment.
Time Frame: as for outcome 10
Population: Participants who received at least one dose of study treatment in Phase 1 Dose Escalation and who had an objective response. Participants were grouped according to assigned total daily dose.
Measure: Median (Full Range); unit: months
Arm/Group | Phase 1 Dose Escalation: Enasidenib 50 mg | Phase 1 Dose Escalation: Enasidenib 60 mg | Phase 1 Dose Escalation: Enasidenib 75 mg | Phase 1 Dose Escalation: Enasidenib 100 mg | Phase 1 Dose Escalation: Enasidenib 150 mg | Phase 1 Dose Escalation: Enasidenib 200 mg | Phase 1 Dose Escalation: Enasidenib 300 mg | Phase 1 Dose Escalation: Enasidenib 450 mg | Phase 1 Dose Escalation: Enasidenib 650 mg
Number analyzed (Participants) | 3 | 3 | 1 | 13 | 6 | 11 | 5 | 3 | 5
months | 4.2 [3.8 to 5.6] | 2.9 [1.0 to 3.8] | 0.9 [0.9 to 0.9] | 2.0 [0.6 to 9.2] | 3.8 [0.6 to 9.7] | 1.9 [0.5 to 5.7] | 3.8 [2.1 to 7.5] | 3.7 [0.5 to 3.8] | 1.9 [0.5 to 3.8]

32. Secondary Outcome: Phase 1 Dose Expansion: Time to Best Response
Description: as for outcome 31
Time Frame: Response assessments were performed every 28 days through Month 12 and every 56 days thereafter until the end of treatment; median duration of treatment exposure in Part 1 Dose Expansion was 5.2 months (range 0.5 to 32.8 months).
Population: Participants who received at least one dose of study treatment in Phase 1 Dose Expansion who had an objective response.
Measure: Median (Full Range); unit: months
Arm/Group | Phase 1 Dose Expansion Arm 1: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 2: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 3: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 4: Enasidenib 100 mg QD
Number analyzed (Participants) | 23 | 5 | 9 | 12
months | 3.7 [0.9 to 11.2] | 3.7 [0.9 to 5.5] | 3.7 [1.8 to 12.9] | 4.6 [0.6 to 14.7]

33. Secondary Outcome: Phase 2 Dose Expansion: Time to Best Response
Description: Time to best response is defined as the time from the date of the first dose to the date of the first occurrence of best response according to the following hierarchical order: CR, CRi/CRp, PR, or MLFS based on the 2003 revised IWG criteria for AML per investigator assessment.
Time Frame: as for outcome 4
Population: as for outcome 17
Measure: Median (Full Range); unit: months
Arm/Group | Phase 2: Enasidenib 100 mg QD
Number analyzed (Participants) | 39
months | 3.7 [0.9 to 12.8]

34. Secondary Outcome: Phase 1 Dose Escalation: Time to Complete Response by Total Daily Dose
Description: Time to complete response is defined as the time from the date of the first dose to the date of the first complete response based on the 2003 revised IWG criteria for AML and 2006 modified IWG criteria for MDS per investigator assessment.
Time Frame: Response assessments were performed every 28 days through Month 12 and every 56 days thereafter until the end of treatment; median duration of treatment exposure in the Phase 1 Dose Escalation phase was 5.0 months (range 0.4 to 34.2 months).
Population: Participants who received at least one dose of study treatment in Phase 1 Dose Escalation with a complete response. Participants were grouped according to assigned total daily dose.
Measure: Median (Full Range); unit: months
Arm/Group | Phase 1 Dose Escalation: Enasidenib 50 mg | Phase 1 Dose Escalation: Enasidenib 60 mg | Phase 1 Dose Escalation: Enasidenib 75 mg | Phase 1 Dose Escalation: Enasidenib 100 mg | Phase 1 Dose Escalation: Enasidenib 150 mg | Phase 1 Dose Escalation: Enasidenib 200 mg | Phase 1 Dose Escalation: Enasidenib 300 mg | Phase 1 Dose Escalation: Enasidenib 450 mg | Phase 1 Dose Escalation: Enasidenib 650 mg
Number analyzed (Participants) | 2 | 1 | 0 | 8 | 2 | 1 | 3 | 2 | 2
months | 4.9 [4.2 to 5.6] | 2.9 [2.9 to 2.9] |  | 3.6 [0.7 to 9.2] | 6.8 [3.8 to 9.7] | 0.6 [0.6 to 0.6] | 4.7 [3.8 to 7.5] | 3.8 [3.7 to 3.8] | 2.1 [0.5 to 3.8]

35. Secondary Outcome: Phase 1 Dose Expansion: Time to Complete Response
Description: as for outcome 34
Time Frame: as for outcome 32
Population: Participants who received at least one dose of study treatment in Phase 1 Dose Expansion who had a complete response.
Measure: Median (Full Range); unit: months
Arm/Group | Phase 1 Dose Expansion Arm 1: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 2: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 3: Enasidenib 100 mg QD | Phase 1 Dose Expansion Arm 4: Enasidenib 100 mg QD
Number analyzed (Participants) | 11 | 0 | 5 | 6
months | 3.7 [1.0 to 11.2] |  | 5.6 [3.4 to 12.9] | 9.4 [1.8 to 14.7]

36. Secondary Outcome: Phase 2 Dose Expansion: Time to Complete Response
Description: Time to complete response is defined as the time from the date of the first dose to the date of the first complete response based on the 2003 revised IWG criteria for AML per investigator assessment.
Time Frame: as for outcome 4
Population: Participants in Phase 2 with R/R AML who received at least one dose of study treatment and who had a complete response.
Measure: Median (Full Range); unit: months
Arm/Group | Phase 2: Enasidenib 100 mg QD
Number analyzed (Participants) | 21
months | 3.7 [0.9 to 12.8]

37. Secondary Outcome: Phase 1: Area Under the Plasma Concentration Time Curve From Time Zero to 8 Hours Postdose (AUC0-8) of Enasidenib After a Single Oral Dose on Day -3
Description: The first 3 participants enrolled in each cohort of the dose escalation phase and the first 15 participants enrolled in each arm of Phase 1 Dose Expansion received a single dose of enasidenib three days prior to starting the 28-day dosing regimen (Day -3) for assessment of enasidenib pharmacokinetics (PK). Plasma enasidenib was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL. Area under the plasma concentration-time curve from time 0 to 8 hours post-dose (AUC0-8) was calculated using the linear trapezoidal rule.
Time Frame: Day -3 prior to the single dose of enasidenib and at 0.5, 1, 2, 3, 4, 6, and 8 hours post-dose.
Population: Participants who received 1 dose of enasidenib on Day -3 with sufficient data to determine PK parameters. Participants who received 2 doses on Day -3 or who received the incorrect dose were excluded. Participants in the Phase 1 Escalation BID and QD cohorts and Phase 1 Expansion cohorts were were grouped by dose for Day -3 analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Enasidenib 30 mg: Participants received a single oral dose of enasidenib 30 mg on Day -3.
- Enasidenib 50 mg: Participants received a single oral dose of enasidenib 50 mg on Day -3.
- Enasidenib 75 mg: Participants received a single oral dose of enasidenib 75 mg on Day -3.
- Enasidenib 100 mg: Participants received a single oral dose of enasidenib 100 mg on Day -3.
- Enasidenib 150 mg: Participants received a single oral dose of enasidenib 150 mg on Day -3.
- Enasidenib 200 mg: Participants received a single oral dose of enasidenib 200 mg on Day -3.
- Enasidenib 300 mg: Participants received a single oral dose of enasidenib 300 mg on Day -3.
- Enasidenib 450 mg: Participants received a single oral dose of enasidenib 450 mg on Day -3.
- Enasidenib 650 mg: Participants received a single oral dose of enasidenib 650 mg on Day -3.
Arm/Group | Enasidenib 30 mg | Enasidenib 50 mg | Enasidenib 75 mg | Enasidenib 100 mg | Enasidenib 150 mg | Enasidenib 200 mg | Enasidenib 300 mg | Enasidenib 450 mg | Enasidenib 650 mg
Number analyzed (Participants) | 4 | 9 | 9 | 58 | 8 | 11 | 6 | 2 | 1
ng*h/mL | 3364 (59.7) | 3020 (58.4) | 5319 (57.0) | 6634 (79.6) | 9397 (32.1) | 11550 (49.2) | 15268 (42.0) | 15039 (NA) — Percent coefficient of variation could not be calculated due to small sample size | 31580 (NA) — Percent coefficient of variation could not be calculated due to small sample size

38. Secondary Outcome: Phase 1: Area Under the Plasma Concentration Time Curve From Time Zero to 10 Hours Postdose (AUC0-10) of Enasidenib After a Single Oral Dose on Day -3
Description: The first 3 participants enrolled in each cohort of the dose escalation phase and the first 15 participants enrolled in each arm of Phase 1 Expansion received a single dose of enasidenib three days prior to starting the 28-day dosing regimen (Day -3). Plasma enasidenib was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL. Area under the plasma concentration-time curve from time 0 to 10 hours post-dose (AUC0-10) was calculated using the linear trapezoidal rule.
Time Frame: Day -3 prior to the single dose of enasidenib and at 0.5, 1, 2, 3, 4, 6, 8, and 10 hours post-dose.
Population: Participants who received 1 dose of enasidenib on Day -3 with sufficient data to determine PK parameters. Participants who received 2 doses on Day -3 or who received the incorrect dose were excluded. Participants in the Phase 1 Escalation BID and QD and Phase 1 Expansion cohorts were were grouped by dose for Day -3 analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Enasidenib 30 mg | Enasidenib 50 mg | Enasidenib 75 mg | Enasidenib 100 mg | Enasidenib 150 mg | Enasidenib 200 mg | Enasidenib 300 mg | Enasidenib 450 mg | Enasidenib 650 mg
Number analyzed (Participants) | 4 | 9 | 9 | 57 | 8 | 11 | 6 | 2 | 1
ng*h/mL | 4120 (61.5) | 3925 (58.4) | 6834 (54.1) | 8616 (76.5) | 11819 (31.3) | 14818 (49.2) | 20727 (41.0) | 19961 (NA) — Percent coefficient of variation could not be calculated due to small sample size | 38711 (NA) — Percent coefficient of variation could not be calculated due to small sample size

39. Secondary Outcome: Phase 1: Area Under the Plasma Concentration Time Curve From Time Zero to 24 Hours Postdose (AUC0-24) of Enasidenib After a Single Oral Dose on Day -3
Description: The first 3 participants enrolled in each cohort of the dose escalation phase and the first 15 participants enrolled in each arm of Phase 1 Expansion received a single dose of enasidenib three days prior to starting the 28-day dosing regimen (Day -3). Plasma enasidenib was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL. Area under the plasma concentration-time curve from time 0 to 24 hours post-dose (AUC0-24) was calculated using the linear trapezoidal rule.
Time Frame: Day -3 prior to the single dose of enasidenib and at 0.5, 1, 2, 3, 4, 6, 8, 10, and 24 hours post-dose.
Population: as for outcome 37
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Enasidenib 30 mg | Enasidenib 50 mg | Enasidenib 75 mg | Enasidenib 100 mg | Enasidenib 150 mg | Enasidenib 200 mg | Enasidenib 300 mg | Enasidenib 450 mg | Enasidenib 650 mg
Number analyzed (Participants) | 4 | 9 | 9 | 56 | 8 | 11 | 6 | 2 | 0
ng*h/mL | 8987 (72.1) | 9611 (59.6) | 17330 (50.6) | 21656 (55.6) | 28989 (29.6) | 37703 (48.3) | 58743 (41.5) | 60846 (NA) — Percent coefficient of variation could not be calculated due to small sample size |

40. Secondary Outcome: Phase 1: Area Under the Plasma Concentration Time Curve From Time Zero to 72 Hours Postdose (AUC0-72) of Enasidenib After a Single Oral Dose on Day -3
Description: The first 3 participants enrolled in each cohort of the dose escalation phase and the first 15 participants enrolled in each arm of Phase 1 Expansion received a single dose of enasidenib three days prior to starting the 28-day dosing regimen (Day -3). Plasma enasidenib was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL. Area under the plasma concentration-time curve from time 0 to 72 hours post-dose (AUC0-72) was calculated using the linear trapezoidal rule.
Time Frame: Day -3 prior to the single dose of enasidenib and at 0.5, 1, 2, 3, 4, 6, 8, 10, 24, 48, and 72 hours post-dose.
Population: as for outcome 37
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Enasidenib 30 mg | Enasidenib 50 mg | Enasidenib 75 mg | Enasidenib 100 mg | Enasidenib 150 mg | Enasidenib 200 mg | Enasidenib 300 mg | Enasidenib 450 mg | Enasidenib 650 mg
Number analyzed (Participants) | 3 | 7 | 8 | 51 | 8 | 9 | 4 | 1 | 0
ng*h/mL | 19192 (138.4) | 20598 (79.9) | 37737 (53.9) | 58670 (59.5) | 76820 (31.2) | 95217 (57.2) | 160083 (12.0) | 244130 (NA) — Percent coefficient of variation could not be calculated due to small sample size |

41. Secondary Outcome: Phase 1: Area Under the Plasma Concentration Time Curve From Time Zero to the Last Quantifiable Concentration (AUC0-t) of Enasidenib After a Single Oral Dose on Day -3
Description: The first 3 participants enrolled in each cohort of the dose escalation phase and the first 15 participants enrolled in each arm of Phase 1 Expansion received a single dose of enasidenib three days prior to starting the 28-day dosing regimen (Day -3). Plasma enasidenib was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL. Area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration (AUC0-t) was calculated using the linear trapezoidal rule.
Time Frame: Day -3 prior to the single dose of enasidenib and at 0.5, 1, 2, 3, 4, 6, 8, 10, 24, 48, and 72 hours post-dose.
Population: as for outcome 37
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Enasidenib 30 mg | Enasidenib 50 mg | Enasidenib 75 mg | Enasidenib 100 mg | Enasidenib 150 mg | Enasidenib 200 mg | Enasidenib 300 mg | Enasidenib 450 mg | Enasidenib 650 mg
Number analyzed (Participants) | 4 | 9 | 9 | 58 | 8 | 11 | 6 | 2 | 1
ng*h/mL | 17575 (105.1) | 19975 (68.6) | 39345 (51.9) | 53018 (74.2) | 76820 (31.2) | 95959 (50.5) | 134094 (32.6) | 157042 (NA) — Percent coefficient of variation could not be calculated due to small sample size | 38711 (NA) — Percent coefficient of variation could not be calculated due to small sample size

42. Secondary Outcome: Phase 1: Maximum Concentration of Enasidenib After a Single Oral Dose on Day -3
Description: The first 3 participants enrolled in each cohort of the dose escalation phase and the first 15 participants enrolled in each arm of Phase 1 Expansion received a single dose of enasidenib three days prior to starting the 28-day dosing regimen (Day -3). Plasma enasidenib was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL.
Time Frame: Day -3 prior to the single dose of enasidenib and at 0.5, 1, 2, 3, 4, 6, 8, 10, 24, 48, and 72 hours post-dose.
Population: as for outcome 37
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Enasidenib 30 mg | Enasidenib 50 mg | Enasidenib 75 mg | Enasidenib 100 mg | Enasidenib 150 mg | Enasidenib 200 mg | Enasidenib 300 mg | Enasidenib 450 mg | Enasidenib 650 mg
Number analyzed (Participants) | 4 | 9 | 9 | 58 | 8 | 11 | 6 | 2 | 1
ng/mL | 569 (45.6) | 545 (64.0) | 1084 (51.6) | 1279 (56.1) | 1624 (29.5) | 2082 (46.5) | 3358 (43.1) | 3031 (NA) — Percent coefficient of variation could not be calculated due to small sample size | 4670 (NA) — Percent coefficient of variation could not be calculated due to small sample size

43. Secondary Outcome: Phase 1: Time to Maximum Concentration (Tmax) of Enasidenib After a Single Oral Dose on Day -3
Description: as for outcome 42
Time Frame: Day -3 prior to the single dose of enasidenib and at 0.5, 1, 2, 3, 4, 6, 8, 10, 24, 48, and 72 hours post-dose.
Population: as for outcome 37
Measure: Median (Full Range); unit: hours
Arm/Group | Enasidenib 30 mg | Enasidenib 50 mg | Enasidenib 75 mg | Enasidenib 100 mg | Enasidenib 150 mg | Enasidenib 200 mg | Enasidenib 300 mg | Enasidenib 450 mg | Enasidenib 650 mg
Number analyzed (Participants) | 4 | 9 | 9 | 58 | 8 | 11 | 6 | 2 | 1
hours | 1.59 [1.00 to 4.08] | 5.83 [1.92 to 24.25] | 3.00 [1.13 to 21.42] | 4.00 [0.67 to 71.97] | 3.98 [2.00 to 24.00] | 4.08 [1.00 to 48.55] | 8.89 [2.95 to 72.17] | 18.61 [13.33 to 23.88] | 6.17 [6.17 to 6.17]

44. Secondary Outcome: Phase 1: Apparent Terminal Phase Half-life (t½) of Enasidenib After a Single Oral Dose on Day -3
Description: The first 3 participants enrolled in each cohort of the dose escalation phase and the first 15 participants enrolled in each arm of Phase 1 Expansion received a single dose of enasidenib three days prior to starting the 28-day dosing regimen (Day -3). Plasma enasidenib was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL. T1/2 was not calculated when the terminal elimination rate constant (λz) was not estimable.
Time Frame: Day -3 prior to the single dose of enasidenib and at 0.5, 1, 2, 3, 4, 6, 8, 10, 24, 48, and 72 hours post-dose.
Population: as for outcome 38
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Enasidenib 30 mg | Enasidenib 50 mg | Enasidenib 75 mg | Enasidenib 100 mg | Enasidenib 150 mg | Enasidenib 200 mg | Enasidenib 300 mg | Enasidenib 450 mg | Enasidenib 650 mg
Number analyzed (Participants) | 3 | 8 | 7 | 29 | 5 | 3 | 2 | 0 | 0
hours | 33.2 (124.6) | 36.8 (57.3) | 52.6 (109.5) | 65.9 (86.5) | 96.2 (60.1) | 73.8 (18.8) | 91.3 (NA) — Percent coefficient of variation could not be calculated due to small sample size |  |

45. Secondary Outcome: Phase 1: AUC From Time Zero to 8 Hours Postdose (AUC0-8) of Enasidenib After Multiple Oral Doses
Description: Plasma enasidenib was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL. Area under the plasma concentration-time curve from time 0 to 8 hours post-dose (AUC0-8) was calculated using the linear trapezoidal rule.
Time Frame: Cycle 2 Day 1 at predose and 0.5, 1, 2, 3, 4, 6, and 8 hours post-dose.
Population: Participants who received enasidenib on Cycle 2, Day 1 with sufficient data to determine PK parameters. Participants who took less than 80% of their planned continuous dosing regimen were excluded from the analysis. Participants in the Phase 1 Escalation and Expansion Enasidenib 100 mg QD cohorts were combined for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Enasidenib 30 mg BID: Participants received enasidenib 30 mg tablets BID on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Enasidenib 50 mg BID: Participants received enasidenib 50 mg tablets BID on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Enasidenib 75 mg BID: Participants received enasidenib 75 mg tablets BID on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Enasidenib 100 mg BID: Participants received enasidenib 100 mg tablets BID on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity
- Enasidenib 150 mg BID: Participants received enasidenib 150 mg tablets BID on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Enasidenib 50 mg QD: Participants received enasidenib 50 mg tablets every day (QD) on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
Arm/Group | Enasidenib 30 mg BID | Enasidenib 50 mg BID | Enasidenib 75 mg BID | Enasidenib 100 mg BID | Enasidenib 150 mg BID | Enasidenib 50 mg QD | Phase 1 Dose Escalation: Enasidenib 75 mg QD | Phase 1 Dose Escalation: Enasidenib 100 mg QD | Phase 1 Dose Escalation: Enasidenib 150 mg QD | Phase 1 Dose Escalation: Enasidenib 200 mg QD | Phase 1 Dose Escalation: Enasidenib 300 mg QD | Phase 1 Dose Escalation: Enasidenib 450 mg QD | Phase 1 Dose Escalation: Enasidenib 650 mg QD
Number analyzed (Participants) | 4 | 7 | 5 | 4 | 4 | 5 | 4 | 102 | 5 | 11 | 7 | 5 | 3
ng*h/mL | 34338 (62.5) | 81775 (35.2) | 103364 (34.1) | 135649 (31.4) | 162308 (18.0) | 43407 (106.5) | 44360 (57.2) | 83444 (48.9) | 101462 (37.7) | 108404 (53.1) | 105098 (40.9) | 181186 (21.5) | 219708 (14.6)

46. Secondary Outcome: Phase 1: AUC From Time Zero to 10 Hours Postdose (AUC0-10) of Enasidenib After Multiple Oral Doses
Description: Plasma enasidenib was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL. Area under the plasma concentration-time curve from time 0 to 10 hours post-dose (AUC0-10) was calculated using the linear trapezoidal rule.
Time Frame: Cycle 2 Day 1 at predose and 0.5, 1, 2, 3, 4, 6, 8, and 10 hours post-dose.
Population: as for outcome 45
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Enasidenib 30 mg BID | Enasidenib 50 mg BID | Enasidenib 75 mg BID | Enasidenib 100 mg BID | Enasidenib 150 mg BID | Enasidenib 50 mg QD | Phase 1 Dose Escalation: Enasidenib 75 mg QD | Phase 1 Dose Escalation: Enasidenib 100 mg QD | Phase 1 Dose Escalation: Enasidenib 150 mg QD | Phase 1 Dose Escalation: Enasidenib 200 mg QD | Phase 1 Dose Escalation: Enasidenib 300 mg QD | Phase 1 Dose Escalation: Enasidenib 450 mg QD | Phase 1 Dose Escalation: Enasidenib 650 mg QD
Number analyzed (Participants) | 4 | 7 | 5 | 4 | 4 | 4 | 4 | 94 | 5 | 11 | 7 | 3 | 2
ng*h/mL | 41108 (63.2) | 99954 (35.1) | 126765 (34.6) | 174409 (32.0) | 200661 (18.9) | 61226 (117.0) | 53067 (50.1) | 104824 (47.6) | 126237 (37.8) | 132718 (52.0) | 131523 (43.0) | 199749 (24.0) | 269750 (NA) — Percent coefficient of variation could not be calculated due to small sample size

47. Secondary Outcome: Phase 1: AUC From Time Zero to the Last Quantifiable Concentration (AUC0-t) of Enasidenib After Multiple Oral Doses
Description: Plasma enasidenib was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL. Area under the plasma concentration-time curve from time 0 to the last quantifiable concentration (AUC0-t) was calculated using the linear trapezoidal rule.
Time Frame: Cycle 2 Day 1 at predose and 0.5, 1, 2, 3, 4, 6, 8, and 10 hours post-dose.
Population: as for outcome 45
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Enasidenib 30 mg BID | Enasidenib 50 mg BID | Enasidenib 75 mg BID | Enasidenib 100 mg BID | Enasidenib 150 mg BID | Enasidenib 50 mg QD | Phase 1 Dose Escalation: Enasidenib 75 mg QD | Phase 1 Dose Escalation: Enasidenib 100 mg QD | Phase 1 Dose Escalation: Enasidenib 150 mg QD | Phase 1 Dose Escalation: Enasidenib 200 mg QD | Phase 1 Dose Escalation: Enasidenib 300 mg QD | Phase 1 Dose Escalation: Enasidenib 450 mg QD | Phase 1 Dose Escalation: Enasidenib 650 mg QD
Number analyzed (Participants) | 4 | 7 | 5 | 4 | 4 | 5 | 4 | 107 | 5 | 11 | 7 | 5 | 3
ng*h/mL | 41108 (63.2) | 99954 (35.1) | 126765 (34.6) | 174409 (32.0) | 200661 (18.9) | 51273 (111.1) | 53067 (50.1) | 100119 (49.7) | 126237 (37.8) | 132718 (52.0) | 131523 (43.0) | 202702 (17.8) | 256155 (16.0)

48. Secondary Outcome: Phase 1: Maximum Concentration (Cmax) of Enasidenib After Multiple Oral Doses
Description: Plasma enasidenib was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL.
Time Frame: Cycle 2 Day 1 at predose and 0.5, 1, 2, 3, 4, 6, 8, and 10 hours post-dose.
Population: as for outcome 45
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Enasidenib 30 mg BID | Enasidenib 50 mg BID | Enasidenib 75 mg BID | Enasidenib 100 mg BID | Enasidenib 150 mg BID | Enasidenib 50 mg QD | Phase 1 Dose Escalation: Enasidenib 75 mg QD | Phase 1 Dose Escalation: Enasidenib 100 mg QD | Phase 1 Dose Escalation: Enasidenib 150 mg QD | Phase 1 Dose Escalation: Enasidenib 200 mg QD | Phase 1 Dose Escalation: Enasidenib 300 mg QD | Phase 1 Dose Escalation: Enasidenib 450 mg QD | Phase 1 Dose Escalation: Enasidenib 650 mg QD
Number analyzed (Participants) | 4 | 7 | 5 | 4 | 4 | 5 | 4 | 107 | 5 | 11 | 7 | 5 | 3
ng/mL | 5300 (71.9) | 12538 (39.2) | 15860 (34.5) | 23962 (25.3) | 26715 (24.7) | 6543 (124.9) | 6922 (64.2) | 13012 (46.5) | 15734 (38.6) | 17990 (64.0) | 18505 (42.4) | 28049 (23.4) | 35269 (10.7)

49. Secondary Outcome: Phase 1: Time to Maximum Concentration (Tmax) of Enasidenib After Multiple Oral Doses
Description: as for outcome 48
Time Frame: Cycle 2 Day 1 at predose and 0.5, 1, 2, 3, 4, 6, 8, and 10 hours post-dose.
Population: as for outcome 45
Measure: Median (Full Range); unit: hours
Arm/Group | Enasidenib 30 mg BID | Enasidenib 50 mg BID | Enasidenib 75 mg BID | Enasidenib 100 mg BID | Enasidenib 150 mg BID | Enasidenib 50 mg QD | Phase 1 Dose Escalation: Enasidenib 75 mg QD | Phase 1 Dose Escalation: Enasidenib 100 mg QD | Phase 1 Dose Escalation: Enasidenib 150 mg QD | Phase 1 Dose Escalation: Enasidenib 200 mg QD | Phase 1 Dose Escalation: Enasidenib 300 mg QD | Phase 1 Dose Escalation: Enasidenib 450 mg QD | Phase 1 Dose Escalation: Enasidenib 650 mg QD
Number analyzed (Participants) | 4 | 7 | 5 | 4 | 4 | 5 | 4 | 107 | 5 | 11 | 7 | 5 | 3
hours | 0.50 [0.00 to 3.92] | 2.00 [0.50 to 9.83] | 0.50 [0.00 to 1.00] | 4.47 [0.48 to 9.83] | 1.54 [1.00 to 9.83] | 3.02 [0.00 to 10.00] | 4.04 [1.00 to 10.08] | 1.02 [0.00 to 10.00] | 2.13 [0.70 to 9.83] | 1.02 [0.00 to 8.00] | 5.98 [0.00 to 9.95] | 4.08 [0.97 to 6.00] | 2.00 [1.95 to 3.00]

50. Secondary Outcome: Phase 2: Area Under the Plasma Concentration Time Curve From Time Zero to 8 Hours Postdose (AUC0-8) of Enasidenib After Single and Multiple Oral Doses
Description: Plasma enasidenib was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL. Area under the plasma concentration-time curve from time 0 to 8 hours post-dose (AUC0-8) of enasidenib was calculated using the linear trapezoidal rule.
Time Frame: Cycle 1 Day 1 and Cycle 2 Day 1 at predose and 2, 4, 6, and 8 hours post-dose.
Population: Participants who received enasidenib on Cycle 1 Day 1 or Cycle 2 Day 1 with sufficient data to determine PK parameters. Participants who took less than 80% of their planned continuous dosing regimen were excluded from the analysis of Cycle 2, Day 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Phase 2: Enasidenib 100 mg QD
Number analyzed (Participants) | 89
ng*h/mL
  Cycle 1, Day 1 | 8134 (49.3)
  Cycle 2, Day 1: number analyzed (Participants) | 63
  Cycle 2, Day 1 | 86505 (44.4)

51. Secondary Outcome: Phase 2: Area Under the Plasma Concentration Time Curve From Time Zero to 24 Hours Postdose (AUC 0-24) of Enasidenib After Single and Multiple Oral Doses
Description: Plasma enasidenib was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL. Area under the plasma concentration-time curve from time 0 to 24 hours post-dose (AUC0-24) was calculated using the linear trapezoidal rule.
Time Frame: Cycle 1 Day 1 and Cycle 2 Day 1 at predose and 2, 4, 6, 8, and 24 hours post-dose.
Population: Participants who received enasidenib on Cycle 1 Day 1 or Cycle 2 Day 1 with sufficient data to determine PK parameters. Participants who took less than 80% of their planned continuous dosing regimen were excluded from the analysis of Cycle 2 Day 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Phase 2: Enasidenib 100 mg QD
Number analyzed (Participants) | 58
ng*h/mL
  Cycle 1, Day 1 | 27889 (46.7)
  Cycle 2, Day 1: number analyzed (Participants) | 48
  Cycle 2, Day 1 | 263131 (42.7)

52. Secondary Outcome: Phase 2: Area Under the Plasma Concentration Time Curve From Time Zero to the Last Quantifiable Concentration (AUC0-t) of Enasidenib After Single and Multiple Oral Doses
Description: as for outcome 47
Time Frame: Cycle 1 Day 1 and Cycle 2 Day 1 at predose and 2, 4, 6, 8, and 24 hours post-dose.
Population: as for outcome 51
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Phase 2: Enasidenib 100 mg QD
Number analyzed (Participants) | 92
ng*h/mL
  Cycle 1, Day 1 | 17447 (88.6)
  Cycle 2, Day 1: number analyzed (Participants) | 69
  Cycle 2, Day 1 | 185566 (75.5)

53. Secondary Outcome: Phase 2: Maximum Concentration (Cmax) of Enasidenib After Single and Multiple Oral Doses
Description: as for outcome 48
Time Frame: Cycle 1 Day 1 and Cycle 2 Day 1 at predose and 2, 4, 6, 8, and 24 hours post-dose.
Population: as for outcome 51
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 2: Enasidenib 100 mg QD
Number analyzed (Participants) | 92
ng/mL
  Cycle 1, Day 1 | 1522 (45.1)
  Cycle 2, Day 1: number analyzed (Participants) | 69
  Cycle 2, Day 1 | 13126 (42.4)

54. Secondary Outcome: Phase 2: Time to Maximum Concentration (Tmax) of Enasidenib After Single and Multiple Oral Doses
Description: as for outcome 48
Time Frame: Cycle 1 Day 1 and Cycle 2 Day 1 at predose and 2, 4, 6, 8, and 24 hours post-dose.
Population: as for outcome 51
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 2: Enasidenib 100 mg QD
Number analyzed (Participants) | 92
hours
  Cycle 1, Day 1 | 4.04 [1.83 to 27.75]
  Cycle 2, Day 1: number analyzed (Participants) | 69
  Cycle 2, Day 1 | 2.08 [0.00 to 23.92]

55. Secondary Outcome: Phase 2: Apparent Terminal Phase Half-life (t1/2) of Enasidenib After Single and Multiple Oral Doses
Description: as for outcome 48
Time Frame: Cycle 1 Day 1 and Cycle 2 Day 1 at predose and 2, 4, 6, 8, and 24 hours post-dose.
Population: Participants who received enasidenib on Cycle 1 Day 1 or Cycle 2 Day 1 with sufficient data to determine PK parameters. Participants who took less than 80% of their planned continuous dosing regimen were excluded from the analysis of Cycle 2 Day 1. t1/2 was not calculated when the terminal elimination rate constant (λz) was not estimable.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Phase 2: Enasidenib 100 mg QD
Number analyzed (Participants) | 19
hours
  Cycle 1, Day 1 | 38.3 (81.7)
  Cycle 2, Day 1: number analyzed (Participants) | 0

56. Secondary Outcome: Phase 1: AUC From Time Zero to 8 Hours Postdose (AUC0-8) of AGI-16903 After a Single Oral Dose of Enasidenib on Day -3
Description: The first 3 participants enrolled in each cohort of the dose escalation phase and the first 15 participants enrolled in each arm of Phase 1 Expansion received a single dose of enasidenib three days prior to starting the 28-day dosing regimen (Day -3). AGI-16903 is a primary metabolite of enasidenib. Plasma AGI-16903 was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL. Area under the plasma concentration-time curve from time 0 to hour 8 post-dose (AUC 0-8) was calculated using the linear trapezoidal rule.
Time Frame: Day -3 prior to the single dose of enasidenib and at 0.5, 1, 2, 3, 4, 6, and 8 hours post-dose.
Population: Participants who received 1 dose of enasidenib on Day -3 with sufficient data to determine PK parameters. Participants who received 2 doses on Day -3 or who received the incorrect dose were excluded. Participants in the Phase 1 Escalation and Expansion cohorts were were grouped by dose for Day -3 analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Enasidenib 30 mg | Enasidenib 50 mg | Enasidenib 75 mg | Enasidenib 100 mg | Enasidenib 150 mg | Enasidenib 200 mg | Enasidenib 300 mg | Enasidenib 450 mg | Enasidenib 650 mg
Number analyzed (Participants) | 4 | 9 | 9 | 55 | 8 | 11 | 6 | 2 | 1
ng*h/mL | 122 (83.6) | 187 (134.4) | 276 (80.6) | 276 (104.1) | 558 (70.3) | 530 (91.1) | 526 (58.8) | 384 (NA) — Percent coefficient of variation could not be calculated due to small sample size | 1470 (NA) — Percent coefficient of variation could not be calculated due to small sample size

57. Secondary Outcome: Phase 1: AUC From Time Zero to 10 Hours Postdose (AUC0-10) of AGI-16903 After a Single Oral Dose of Enasidenib on Day -3
Description: The first 3 participants enrolled in each cohort of the dose escalation phase and the first 15 participants enrolled in each arm of Phase 1 Expansion received a single dose of enasidenib three days prior to starting the 28-day dosing regimen (Day -3). AGI-16903 is a primary metabolite of enasidenib. Plasma AGI-16903 was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL. Area under the plasma concentration-time curve from time 0 to 10 hours post-dose (AUC0-10) was calculated using the linear trapezoidal rule.
Time Frame: Day -3 prior to the single dose of enasidenib and at 0.5, 1, 2, 3, 4, 6, 8, and 10 hours post-dose.
Population: as for outcome 38
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Enasidenib 30 mg | Enasidenib 50 mg | Enasidenib 75 mg | Enasidenib 100 mg | Enasidenib 150 mg | Enasidenib 200 mg | Enasidenib 300 mg | Enasidenib 450 mg | Enasidenib 650 mg
Number analyzed (Participants) | 4 | 9 | 9 | 54 | 8 | 11 | 6 | 2 | 1
ng*h/mL | 162 (80.4) | 258 (135.1) | 383 (72.3) | 379 (99.3) | 735 (65.1) | 716 (86.8) | 757 (57.5) | 548 (NA) — Percent coefficient of variation could not be calculated due to small sample size | 1893 (NA) — Percent coefficient of variation could not be calculated due to small sample size

58. Secondary Outcome: Phase 1: AUC From Time Zero to 24 Hours Postdose (AUC0-24) of AGI-16903 After a Single Oral Dose of Enasidenib on Day -3
Description: The first 3 participants enrolled in each cohort of the dose escalation phase and the first 15 participants enrolled in each arm of Phase 1 Expansion received a single dose of enasidenib three days prior to starting the 28-day dosing regimen (Day -3). AGI-16903 is a primary metabolite of enasidenib. Plasma AGI-16903 was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL. Area under the plasma concentration-time curve from time 0 to 24 hours post-dose (AUC0-24) was calculated using the linear trapezoidal rule.
Time Frame: Day -3 prior to the single dose of enasidenib and at 0.5, 1, 2, 3, 4, 6, 8, 10, and 24 hours post-dose.
Population: as for outcome 37
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Enasidenib 30 mg | Enasidenib 50 mg | Enasidenib 75 mg | Enasidenib 100 mg | Enasidenib 150 mg | Enasidenib 200 mg | Enasidenib 300 mg | Enasidenib 450 mg | Enasidenib 650 mg
Number analyzed (Participants) | 4 | 9 | 9 | 53 | 8 | 11 | 6 | 2 | 0
ng*h/mL | 474 (80.4) | 777 (111.7) | 1238 (54.4) | 1222 (71.4) | 2128 (54.2) | 2159 (75.4) | 2477 (51.5) | 2274 (NA) — Percent coefficient of variation could not be calculated due to small sample size |

59. Secondary Outcome: Phase 1: AUC From Time Zero to 72 Hours Postdose (AUC0-72) of AGI-16903 After a Single Oral Dose of Enasidenib on Day -3
Description: The first 3 participants enrolled in each cohort of the dose escalation phase and the first 15 participants enrolled in each arm of Phase 1 Expansion received a single dose of enasidenib three days prior to starting the 28-day dosing regimen (Day -3). AGI-16903 is a primary metabolite of enasidenib. Plasma AGI-16903 was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL. Area under the plasma concentration-time curve from time 0 to 72 hours post-dose (AUC0-72) was calculated using the linear trapezoidal rule.
Time Frame: Day -3 prior to the single dose of enasidenib and at 0.5, 1, 2, 3, 4, 6, 8, 10, 24, 48, and 72 hours post-dose.
Population: as for outcome 37
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Enasidenib 30 mg | Enasidenib 50 mg | Enasidenib 75 mg | Enasidenib 100 mg | Enasidenib 150 mg | Enasidenib 200 mg | Enasidenib 300 mg | Enasidenib 450 mg | Enasidenib 650 mg
Number analyzed (Participants) | 4 | 7 | 8 | 48 | 8 | 9 | 4 | 1 | 0
ng*h/mL | 1403 (93.7) | 2121 (104.8) | 3427 (40.9) | 4283 (58.0) | 7188 (43.6) | 7634 (66.2) | 10673 (29.8) | 17591 (NA) — Percent coefficient of variation could not be calculated due to small sample size |

60. Secondary Outcome: Phase 1: AUC From Time Zero to the Last Quantifiable Concentration (AUC0-t) of AGI-16903 After a Single Oral Dose of Enasidenib on Day -3
Description: The first 3 participants enrolled in each cohort of the dose escalation phase and the first 15 participants enrolled in each arm of Phase 1 Expansion received a single dose of enasidenib three days prior to starting the 28-day dosing regimen (Day -3). AGI-16903 is a primary metabolite of enasidenib. Plasma AGI-16903 was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL. Area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration (AUC0-t) was calculated using the linear trapezoidal rule.
Time Frame: Day -3 prior to the single dose of enasidenib and at 0.5, 1, 2, 3, 4, 6, 8, 10, 24, 48, and 72 hours post-dose.
Population: as for outcome 37
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Enasidenib 30 mg | Enasidenib 50 mg | Enasidenib 75 mg | Enasidenib 100 mg | Enasidenib 150 mg | Enasidenib 200 mg | Enasidenib 300 mg | Enasidenib 450 mg | Enasidenib 650 mg
Number analyzed (Participants) | 4 | 9 | 9 | 55 | 8 | 11 | 6 | 2 | 1
ng*h/mL | 1403 (93.7) | 2101 (86.2) | 3560 (40.0) | 3764 (83.8) | 7188 (43.6) | 7070 (62.0) | 6531 (93.9) | 8035 (NA) — Percent coefficient of variation could not be calculated due to small sample size | 1893 (NA) — Percent coefficient of variation could not be calculated due to small sample size

61. Secondary Outcome: Phase 1: Maximum Concentration of AGI-16903 After a Single Oral Dose of Enasidenib on Day -3
Description: The first 3 participants enrolled in each cohort of the dose escalation phase and the first 15 participants enrolled in each arm of Phase 1 Expansion received a single dose of enasidenib three days prior to starting the 28-day dosing regimen (Day -3). AGI-16903 is a primary metabolite of enasidenib. Plasma AGI-16903 was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL.
Time Frame: Day -3 prior to the single dose of enasidenib and at 0.5, 1, 2, 3, 4, 6, 8, 10, 24, 48, and 72 hours post-dose.
Population: as for outcome 37
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Enasidenib 30 mg | Enasidenib 50 mg | Enasidenib 75 mg | Enasidenib 100 mg | Enasidenib 150 mg | Enasidenib 200 mg | Enasidenib 300 mg | Enasidenib 450 mg | Enasidenib 650 mg
Number analyzed (Participants) | 4 | 9 | 9 | 55 | 8 | 11 | 6 | 2 | 1
ng/mL | 29 (89.3) | 47 (68.3) | 74 (52.3) | 79 (60.6) | 126 (39.4) | 138 (47.4) | 151 (52.4) | 188 (NA) — Percent coefficient of variation could not be calculated due to small sample size | 242 (NA) — Percent coefficient of variation could not be calculated due to small sample size

62. Secondary Outcome: Phase 1: Time to Maximum Concentration (Tmax) of AGI-16903 After a Single Oral Dose of Enasidenib on Day -3
Description: as for outcome 61
Time Frame: Day -3 prior to the single dose of enasidenib and at 0.5, 1, 2, 3, 4, 6, 8, 10, 24, 48, and 72 hours post-dose.
Population: as for outcome 37
Measure: Median (Full Range); unit: hours
Arm/Group | Enasidenib 30 mg | Enasidenib 50 mg | Enasidenib 75 mg | Enasidenib 100 mg | Enasidenib 150 mg | Enasidenib 200 mg | Enasidenib 300 mg | Enasidenib 450 mg | Enasidenib 650 mg
Number analyzed (Participants) | 4 | 9 | 9 | 55 | 8 | 11 | 6 | 2 | 1
hours | 36.38 [3.00 to 70.42] | 10.00 [1.92 to 69.50] | 10.00 [3.00 to 71.00] | 48.00 [3.00 to 74.42] | 24.12 [6.20 to 72.10] | 47.33 [1.98 to 72.82] | 48.10 [7.95 to 72.17] | 59.88 [48.25 to 71.50] | 6.17 [6.17 to 6.17]

63. Secondary Outcome: Phase 1: Apparent Terminal Phase Half-life (t½) of AGI-16903 After a Single Oral Dose of Enasidenib on Day -3
Description: The first 3 participants enrolled in each cohort of the dose escalation phase and the first 15 participants enrolled in each arm of Phase 1 Expansion received a single dose of enasidenib three days prior to starting the 28-day dosing regimen (Day -3). AGI-16903 is a primary metabolite of enasidenib. Plasma AGI-16903 was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL. t1/2 was not calculated when the terminal elimination rate constant (λz) was not estimable.
Time Frame: Day -3 prior to the single dose of enasidenib and at 0.5, 1, 2, 3, 4, 6, 8, 10, 24, 48, and 72 hours post-dose.
Population: as for outcome 37
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Enasidenib 30 mg | Enasidenib 50 mg | Enasidenib 75 mg | Enasidenib 100 mg | Enasidenib 150 mg | Enasidenib 200 mg | Enasidenib 300 mg | Enasidenib 450 mg | Enasidenib 650 mg
Number analyzed (Participants) | 1 | 4 | 2 | 7 | 1 | 0 | 0 | 0 | 0
hours | 18.9 (NA) — Percent coefficient of variation could not be calculated due to small sample size | 46.9 (125.7) | 29.0 (NA) — Percent coefficient of variation could not be calculated due to small sample size | 69.2 (161.0) | 106.4 (NA) — Percent coefficient of variation could not be calculated due to small sample size |  |  |  |

64. Secondary Outcome: Phase 1: AUC From Time Zero to 8 Hours Postdose (AUC0-8) of AGI-16903 After Multiple Oral Doses of Enasidenib
Description: AGI-16903 is a primary metabolite of enasidenib. Plasma AGI-16903 was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL. Area under the plasma concentration-time curve from time 0 to 8 hours post-dose (AUC0-8) was calculated using the linear trapezoidal rule.
Time Frame: Cycle 2 Day 1 at predose and 0.5, 1, 2, 3, 4, 6, and 8 hours post-dose.
Population: as for outcome 45
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Enasidenib 30 mg BID | Enasidenib 50 mg BID | Enasidenib 75 mg BID | Enasidenib 100 mg BID | Enasidenib 150 mg BID | Enasidenib 50 mg QD | Phase 1 Dose Escalation: Enasidenib 75 mg QD | Phase 1 Dose Escalation: Enasidenib 100 mg QD | Phase 1 Dose Escalation: Enasidenib 150 mg QD | Phase 1 Dose Escalation: Enasidenib 200 mg QD | Phase 1 Dose Escalation: Enasidenib 300 mg QD | Phase 1 Dose Escalation: Enasidenib 450 mg QD | Phase 1 Dose Escalation: Enasidenib 650 mg QD
Number analyzed (Participants) | 4 | 7 | 5 | 2 | 4 | 5 | 4 | 102 | 3 | 11 | 7 | 5 | 3
ng*h/mL | 4028 (82.9) | 7656 (47.5) | 7340 (59.8) | 10655 (NA) — Percent coefficient of variation could not be calculated due to small sample size | 16638 (15.7) | 4395 (125.7) | 3281 (87.3) | 7645 (42.7) | 10720 (38.3) | 11579 (47.5) | 9961 (36.0) | 15888 (35.4) | 20480 (36.8)

65. Secondary Outcome: Phase 1: AUC From Time Zero to 10 Hours Postdose (AUC0-10) of AGI-16903 After Multiple Oral Doses of Enasidenib
Description: AGI-16903 is a primary metabolite of enasidenib. Plasma AGI-16903 was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL. Area under the plasma concentration-time curve from time 0 to 10 hours post-dose (AUC0-10) was calculated using the linear trapezoidal rule.
Time Frame: Cycle 2 Day 1 at predose and 0.5, 1, 2, 3, 4, 6, 8, and 10 hours post-dose.
Population: as for outcome 45
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Enasidenib 30 mg BID | Enasidenib 50 mg BID | Enasidenib 75 mg BID | Enasidenib 100 mg BID | Enasidenib 150 mg BID | Enasidenib 50 mg QD | Phase 1 Dose Escalation: Enasidenib 75 mg QD | Phase 1 Dose Escalation: Enasidenib 100 mg QD | Phase 1 Dose Escalation: Enasidenib 150 mg QD | Phase 1 Dose Escalation: Enasidenib 200 mg QD | Phase 1 Dose Escalation: Enasidenib 300 mg QD | Phase 1 Dose Escalation: Enasidenib 450 mg QD | Phase 1 Dose Escalation: Enasidenib 650 mg QD
Number analyzed (Participants) | 4 | 7 | 5 | 2 | 4 | 4 | 4 | 94 | 3 | 11 | 7 | 3 | 2
ng*h/mL | 4830 (82.9) | 9437 (46.8) | 9002 (60.0) | 13463 (NA) — Percent coefficient of variation could not be calculated due to small sample size | 20705 (16.1) | 6502 (132.7) | 3954 (80.6) | 9502 (42.0) | 13263 (40.1) | 14303 (47.2) | 12448 (35.0) | 17963 (18.7) | 22102 (NA) — Percent coefficient of variation could not be calculated due to small sample size

66. Secondary Outcome: Phase 1: AUC From Time Zero to the Last Quantifiable Concentration (AUC0-t) of AGI-16903 After Multiple Oral Doses of Enasidenib
Description: AGI-16903 is a primary metabolite of enasidenib. Plasma AGI-16903 was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL. Area under the plasma concentration-time curve from time 0 to the last quantifiable concentration (AUC0-t) was calculated using the linear trapezoidal rule.
Time Frame: Cycle 2 Day 1 at predose and 0.5, 1, 2, 3, 4, 6, 8, and 10 hours post-dose.
Population: as for outcome 45
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Enasidenib 30 mg BID | Enasidenib 50 mg BID | Enasidenib 75 mg BID | Enasidenib 100 mg BID | Enasidenib 150 mg BID | Enasidenib 50 mg QD | Phase 1 Dose Escalation: Enasidenib 75 mg QD | Phase 1 Dose Escalation: Enasidenib 100 mg QD | Phase 1 Dose Escalation: Enasidenib 150 mg QD | Phase 1 Dose Escalation: Enasidenib 200 mg QD | Phase 1 Dose Escalation: Enasidenib 300 mg QD | Phase 1 Dose Escalation: Enasidenib 450 mg QD | Phase 1 Dose Escalation: Enasidenib 650 mg QD
Number analyzed (Participants) | 4 | 7 | 5 | 2 | 4 | 5 | 4 | 107 | 3 | 11 | 7 | 5 | 3
ng*h/mL | 4830 (82.9) | 9437 (46.8) | 9002 (60.0) | 13463 (NA) — Percent coefficient of variation could not be calculated due to small sample size | 20705 (16.1) | 5181 (133.1) | 3954 (80.6) | 9193 (42.1) | 13263 (40.1) | 14303 (47.2) | 12448 (35.0) | 17846 (33.7) | 24187 (24.4)

67. Secondary Outcome: Phase 1: Maximum Concentration (Cmax) of AGI-16903 After Multiple Oral Doses of Enasidenib
Description: AGI-16903 is a primary metabolite of enasidenib. Plasma AGI-16903 was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL.
Time Frame: Cycle 2 Day 1 at predose and 0.5, 1, 2, 3, 4, 6, 8, and 10 hours post-dose.
Population: as for outcome 45
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Enasidenib 30 mg BID | Enasidenib 50 mg BID | Enasidenib 75 mg BID | Enasidenib 100 mg BID | Enasidenib 150 mg BID | Enasidenib 50 mg QD | Phase 1 Dose Escalation: Enasidenib 75 mg QD | Phase 1 Dose Escalation: Enasidenib 100 mg QD | Phase 1 Dose Escalation: Enasidenib 150 mg QD | Phase 1 Dose Escalation: Enasidenib 200 mg QD | Phase 1 Dose Escalation: Enasidenib 300 mg QD | Phase 1 Dose Escalation: Enasidenib 450 mg QD | Phase 1 Dose Escalation: Enasidenib 650 mg QD
Number analyzed (Participants) | 4 | 7 | 5 | 2 | 4 | 5 | 4 | 107 | 3 | 11 | 7 | 5 | 3
ng/mL | 619 (95.0) | 1149 (54.0) | 1096 (62.8) | 1717 (NA) — Percent coefficient of variation could not be calculated due to small sample size | 2651 (13.6) | 680 (148.1) | 518 (99.8) | 1199 (42.3) | 1640 (30.2) | 1817 (55.0) | 1687 (37.7) | 2415 (33.2) | 3135 (38.8)

68. Secondary Outcome: Phase 1: Time to Maximum Concentration (Tmax) of AGI-16903 After Multiple Oral Doses of Enasidenib
Description: as for outcome 67
Time Frame: Cycle 2 Day 1 at predose and 0.5, 1, 2, 3, 4, 6, 8, and 10 hours post-dose.
Population: as for outcome 45
Measure: Median (Full Range); unit: hours
Arm/Group | Enasidenib 30 mg BID | Enasidenib 50 mg BID | Enasidenib 75 mg BID | Enasidenib 100 mg BID | Enasidenib 150 mg BID | Enasidenib 50 mg QD | Phase 1 Dose Escalation: Enasidenib 75 mg QD | Phase 1 Dose Escalation: Enasidenib 100 mg QD | Phase 1 Dose Escalation: Enasidenib 150 mg QD | Phase 1 Dose Escalation: Enasidenib 200 mg QD | Phase 1 Dose Escalation: Enasidenib 300 mg QD | Phase 1 Dose Escalation: Enasidenib 450 mg QD | Phase 1 Dose Escalation: Enasidenib 650 mg QD
Number analyzed (Participants) | 4 | 7 | 5 | 2 | 4 | 5 | 4 | 107 | 3 | 11 | 7 | 5 | 3
hours | 1.50 [0.00 to 4.17] | 2.00 [1.00 to 10.00] | 0.52 [0.33 to 7.97] | 1.48 [1.00 to 1.97] | 1.54 [1.00 to 8.00] | 2.92 [0.00 to 3.92] | 1.58 [1.00 to 6.08] | 1.00 [0.00 to 10.00] | 4.00 [2.00 to 9.83] | 1.00 [0.00 to 8.00] | 5.98 [0.00 to 9.95] | 2.98 [0.97 to 6.00] | 1.97 [1.95 to 10.00]

69. Secondary Outcome: Phase 2: AUC From Time Zero to 8 Hours Postdose (AUC0-8) of AGI-16903 After Single and Multiple Oral Doses of Enasidenib
Description: as for outcome 64
Time Frame: Cycle 1 Day 1 and Cycle 2 Day 1 at predose and 2, 4, 6, and 8 hours post-dose.
Population: Participants who received enasidenib on Cycle 1, Day 1 or Cycle 2, Day 1 with sufficient data to determine PK parameters. Participants who took less than 80% of their planned continuous dosing regimen were excluded from the analysis of Cycle 2, Day 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Phase 2: Enasidenib 100 mg QD
Number analyzed (Participants) | 88
ng*h/mL
  Cycle 1, Day 1 | 323 (90.8)
  Cycle 2, Day 1: number analyzed (Participants) | 62
  Cycle 2, Day 1 | 7409 (45.3)

70. Secondary Outcome: Phase 2: AUC From Time Zero to 24 Hours Postdose (AUC0-24) of AGI-16903 After Single and Multiple Oral Doses of Enasidenib
Description: AGI-16903 is a primary metabolite of enasidenib. Plasma AGI-16903 was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL. Area under the plasma concentration-time curve from time 0 to 24 hours post-dose (AUC0-24) was calculated using the linear trapezoidal rule.
Time Frame: Cycle 1 Day 1 and Cycle 2 Day 1 at predose and 2, 4, 6, 8, and 24 hours post-dose.
Population: as for outcome 69
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Phase 2: Enasidenib 100 mg QD
Number analyzed (Participants) | 58
ng*h/mL
  Cycle 1, Day 1 | 1482 (63.9)
  Cycle 2, Day 1: number analyzed (Participants) | 48
  Cycle 2, Day 1 | 23963 (43.8)

71. Secondary Outcome: Phase 2: AUC From Time Zero to the Last Quantifiable Concentration (AUC0-t) of AGI-16903 After Single and Multiple Oral Doses of Enasidenib
Description: as for outcome 66
Time Frame: Cycle 1 Day 1 and Cycle 2 Day 1 at predose and 2, 4, 6, 8, and 24 hours post-dose.
Population: as for outcome 69
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Phase 2: Enasidenib 100 mg QD
Number analyzed (Participants) | 91
ng*h/mL
  Cycle 1, Day 1 | 829 (138.1)
  Cycle 2, Day 1: number analyzed (Participants) | 68
  Cycle 2, Day 1 | 16593 (81.8)

72. Secondary Outcome: Phase 2: Maximum Concentration (Cmax) of AGI-16903 After Single and Multiple Oral Doses of Enasidenib
Description: as for outcome 67
Time Frame: Cycle 1 Day 1 and Cycle 2 Day 1 at predose and 2, 4, 6, 8, and 24 hours post-dose.
Population: as for outcome 69
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 2: Enasidenib 100 mg QD
Number analyzed (Participants) | 91
ng/mL
  Cycle 1, Day 1 | 72 (80.8)
  Cycle 2, Day 1: number analyzed (Participants) | 68
  Cycle 2, Day 1 | 1158 (48.5)

73. Secondary Outcome: Phase 2: Time to Maximum Concentration (Tmax) of AGI-16903 After Single and Multiple Oral Doses of Enasidenib
Description: as for outcome 67
Time Frame: Cycle 1 Day 1 and Cycle 2 Day 1 at predose and 2, 4, 6, 8, and 24 hours post-dose.
Population: as for outcome 69
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 2: Enasidenib 100 mg QD
Number analyzed (Participants) | 91
hours
  Cycle 1, Day 1 | 8.00 [2.00 to 29.02]
  Cycle 2, Day 1: number analyzed (Participants) | 68
  Cycle 2, Day 1 | 2.12 [0.00 to 23.92]

74. Secondary Outcome: Phase 2: Apparent Terminal Phase Half-life (t1/2) of AGI-16903 After Single and Multiple Oral Doses of Enasidenib
Description: as for outcome 67
Time Frame: Cycle 1 Day 1 and Cycle 2 Day 1 at predose and 2, 4, 6, 8, and 24 hours post-dose.
Population: Participants who received enasidenib on Cycle 1, Day 1 or Cycle 2, Day 1 with sufficient data to determine PK parameters. Participants who took less than 80% of their planned continuous dosing regimen were excluded from the analysis of Cycle 2, Day 1. T1/2 was not calculated when the terminal elimination rate constant (λz) was not estimable.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Phase 2: Enasidenib 100 mg QD
Number analyzed (Participants) | 4
hours
  Cycle 1, Day 1 | 32.2 (116.9)
  Cycle 2, Day 1: number analyzed (Participants) | 0

75. Secondary Outcome: Phase 1 and 2: AUC From Time Zero to 8 Hours Postdose (AUC0-8) After Single and Multiple Oral Doses of Enasidenib 100 mg QD
Description: The first 3 participants enrolled in each cohort of the dose escalation phase and the first 15 participants enrolled in each arm of Phase 1 Expansion received a single dose of enasidenib three days prior to starting the 28-day dosing regimen (Day -3) for single dose PK analysis, and underwent PK assessments on Cycle 2, Day 1 for multiple dose (steady-state) PK analysis. Participants in Phase 2 underwent PK assessments on Cycle 1, Day 1 for single dose analysis and on Cycle 2, Day 1 for multiple dose (steady-state) analysis. Plasma enasidenib was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL. Area under the plasma concentration-time curve from time 0 to 8 hours post-dose (AUC0-8) was calculated using the linear trapezoidal rule.
Time Frame: Day -3 (Phase 1 only) predose and at 0.5, 1, 2, 3, 4, 6, and 8 hours post-dose or Cycle 1 Day 1 (Phase 2) and Cycle 2 Day 1 (Phase 1 & 2) at predose and 2, 4, 6, and 8 hours post-dose.
Population: Participants who received enasidenib on Day -3 or Cycle 1, Day 1 and Cycle 2, Day 1 with sufficient data to determine PK parameters. Participants who took < 80% of their planned continuous dosing regimen were excluded from the analysis of Cycle 2, Day 1. Participants in Phase 1 and 2 who received enasidenib 100 mg QD are combined for the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Phase 1 and 2: Enasidenib 100 mg QD: Participants in Phase 1 and 2 who received 100 mg enasidenib QD on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
Arm/Group | Phase 1 and 2: Enasidenib 100 mg QD
Number analyzed (Participants) | 165
ng*h/mL
  Day -3 / Cycle 1, Day 1: number analyzed (Participants) | 147
  Day -3 / Cycle 1, Day 1 | 7506 (62.8)
  Cycle 2, Day 1 | 84600 (47.1)

76. Secondary Outcome: Phase 1 and 2: AUC From Time Zero to 24 Hours Postdose (AUC0-24) After Single and Multiple Oral Doses of Enasidenib 100 mg QD
Description: The first 3 participants enrolled in each cohort of the dose escalation phase and the first 15 participants enrolled in each arm of Phase 1 Expansion received a single dose of enasidenib three days prior to starting the 28-day dosing regimen (Day -3) for single dose PK analysis, and underwent PK assessments on Cycle 2, Day 1 for multiple dose (steady-state) PK analysis. Participants in Phase 2 underwent PK assessments on Cycle 1, Day 1 for single dose analysis and on Cycle 2, Day 1 for multiple dose (steady-state) analysis. Plasma enasidenib was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL. Area under the plasma concentration-time curve from time 0 to 24 hours post-dose (AUC0-24) was calculated using the linear trapezoidal rule.
Time Frame: Day -3 (Phase 1 only) predose and at 0.5, 1, 2, 3, 4, 6, 8, 10, and 24 hours post-dose or Cycle 1 Day 1 (Phase 2) and Cycle 2 Day 1 (Phase 1 & 2) at predose and 2, 4, 6, 8, and 24 hours post-dose.
Population: as for outcome 75
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Phase 1 and 2: Enasidenib 100 mg QD
Number analyzed (Participants) | 114
ng*h/mL
  Day -3 / Cycle 1, Day 1 | 24631 (52.9)
  Cycle 2, Day 1: number analyzed (Participants) | 48
  Cycle 2, Day 1 | 263131 (42.7)

77. Secondary Outcome: Phase 1 and 2: Maximum Concentration (Cmax) After Single and Multiple Oral Doses of Enasidenib 100 mg QD
Description: The first 3 participants enrolled in each cohort of the dose escalation phase and the first 15 participants enrolled in each arm of Phase 1 Expansion received a single dose of enasidenib three days prior to starting the 28-day dosing regimen (Day -3) for single dose PK analysis, and underwent PK assessments on Cycle 2, Day 1 for multiple dose (steady-state) PK analysis. Participants in Phase 2 underwent PK assessments on Cycle 1, Day 1 for single dose analysis and on Cycle 2, Day 1 for multiple dose (steady-state) analysis. Plasma enasidenib was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL.
Time Frame: Day -3 (Phase 1 only) predose and at 0.5, 1, 2, 3, 4, 6, 8, 10, 24, 48, and 72 hours post-dose or Cycle 1 Day 1 (Phase 2) and Cycle 2 Day 1 (Phase 1 & 2) at predose and 2, 4, 6, 8, and 24 hours post-dose.
Population: as for outcome 75
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1 and 2: Enasidenib 100 mg QD
Number analyzed (Participants) | 176
ng/mL
  Day -3 / Cycle 1, Day 1: number analyzed (Participants) | 150
  Day -3 / Cycle 1, Day 1 | 1423 (50.2)
  Cycle 2, Day 1 | 13057 (44.8)

78. Secondary Outcome: Phase 1 and 2: Time to Maximum Concentration (Tmax) After Single and Multiple Oral Doses of Enasidenib 100 mg QD
Description: as for outcome 77
Time Frame: as for outcome 77
Population: as for outcome 75
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 1 and 2: Enasidenib 100 mg QD
Number analyzed (Participants) | 176
hours
  Day -3 / Cycle 1, Day 1: number analyzed (Participants) | 150
  Day -3 / Cycle 1, Day 1 | 4.00 [0.67 to 71.97]
  Cycle 2, Day 1 | 2.00 [0.00 to 23.92]

79. Secondary Outcome: Phase 1 and 2: AUC From Time Zero to 8 Hours Postdose (AUC0-8) of AGI-16903 After Single and Multiple Oral Doses of Enasidenib 100 mg QD
Description: The first 3 participants enrolled in each cohort of the dose escalation phase and the first 15 participants enrolled in each arm of Phase 1 Expansion received a single dose of enasidenib three days prior to starting the 28-day dosing regimen (Day -3) for single dose PK analysis, and underwent PK assessments on Cycle 2, Day 1 for multiple dose (steady-state) PK analysis. Participants in Phase 2 underwent PK assessments on Cycle 1, Day 1 for single dose analysis and on Cycle 2, Day 1 for multiple dose (steady-state) analysis. AGI-16903 is a primary metabolite of enasidenib. Plasma AGI-16903 was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL. Area under the plasma concentration-time curve from time 0 to 8 hours post-dose (AUC0-8) was calculated using the linear trapezoidal rule.
Time Frame: as for outcome 75
Population: as for outcome 75
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Phase 1 and 2: Enasidenib 100 mg QD
Number analyzed (Participants) | 164
ng*h/mL
  Day -3 / Cycle 1, Day 1: number analyzed (Participants) | 143
  Day -3 / Cycle 1, Day 1 | 304 (96.0)
  Cycle 2, Day 1 | 7555 (43.6)

80. Secondary Outcome: Phase 1 and 2: AUC From Time Zero to 24 Hours Postdose (AUC0-24) of AGI-16903 After Single and Multiple Oral Doses of Enasidenib 100 mg QD
Description: The first 3 participants enrolled in each cohort of the dose escalation phase and the first 15 participants enrolled in each arm of Phase 1 Expansion received a single dose of enasidenib three days prior to starting the 28-day dosing regimen (Day -3) for single dose PK analysis, and underwent PK assessments on Cycle 2, Day 1 for multiple dose (steady-state) PK analysis. Participants in Phase 2 underwent PK assessments on Cycle 1, Day 1 for single dose analysis and on Cycle 2, Day 1 for multiple dose (steady-state) analysis. AGI-16903 is a primary metabolite of enasidenib. Plasma AGI-16903 was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL. Area under the plasma concentration-time curve from time 0 to 24 hours post-dose (AUC0-24) was calculated using the linear trapezoidal rule.
Time Frame: as for outcome 76
Population: as for outcome 75
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Phase 1 and 2: Enasidenib 100 mg QD
Number analyzed (Participants) | 111
ng*h/mL
  Day -3 / Cycle 1, Day 1 | 1352 (68.2)
  Cycle 2, Day 1: number analyzed (Participants) | 48
  Cycle 2, Day 1 | 23963 (43.8)

81. Secondary Outcome: Phase 1 and 2: Maximum Concentration (Cmax) of AGI-16903 After Single and Multiple Oral Doses of Enasidenib 100 mg QD
Description: The first 3 participants enrolled in each cohort of the dose escalation phase and the first 15 participants enrolled in each arm of Phase 1 Expansion received a single dose of enasidenib three days prior to starting the 28-day dosing regimen (Day -3) for single dose PK analysis, and underwent PK assessments on Cycle 2, Day 1 for multiple dose (steady-state) PK analysis. Participants in Phase 2 underwent PK assessments on Cycle 1, Day 1 for single dose analysis and on Cycle 2, Day 1 for multiple dose (steady-state) analysis. AGI-16903 is a primary metabolite of enasidenib. Plasma AGI-16903 was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL.
Time Frame: as for outcome 77
Population: as for outcome 75
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1 and 2: Enasidenib 100 mg QD
Number analyzed (Participants) | 175
ng/mL
  Day -3 / Cycle 1, Day 1: number analyzed (Participants) | 146
  Day -3 / Cycle 1, Day 1 | 75 (73.3)
  Cycle 2, Day 1 | 1183 (44.7)

82. Secondary Outcome: Phase 1 and 2: Time to Maximum Concentration (Tmax) of AGI-16903 After Single and Multiple Oral Doses of Enasidenib 100 mg QD
Description: as for outcome 81
Time Frame: as for outcome 77
Population: as for outcome 75
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 1 and 2: Enasidenib 100 mg QD
Number analyzed (Participants) | 175
hours
  Day -3 / Cycle 1, Day 1: number analyzed (Participants) | 146
  Day -3 / Cycle 1, Day 1 | 23.44 [2.00 to 74.42]
  Cycle 2, Day 1 | 1.92 [0.00 to 23.92]

83. Secondary Outcome: Phase 1: Percent Change From Baseline for Area Under the Effect Concentration Time Curve From Time 0 to 10 Hours Postdose (%BAUEC0-10) of 2-hydroxyglutarate (2-HG) on Day -3
Description: The first 3 participants enrolled in each cohort of the dose escalation phase and the first 15 participants enrolled in each arm of Phase 1 Expansion received a single dose of enasidenib three days prior to starting the 28-day dosing regimen (Day -3). Plasma 2-HG was measured using qualified LC-MS/MS in order to characterize the pharmacodynamic (PD) effects of enasidenib; the LLOQ was 30.0 ng/mL. Area under the effect concentration time curve from time point zero (predose) up to 10 hours postdose (AUEC0-10) was calculated using the linear trapezoid rule. Percent change from Baseline for AUEC0-10 was calculated as (AUEC0-10 minus [Baseline*Tlast]) / (Baseline*Tlast) * 100, where Tlast corresponded to 10 hours and Baseline was equal to the average of the Screening and Day -3 (predose) 2-HG values. Data reported are the arithmetic mean and relative standard deviation expressed as a percentage.
Time Frame: Screening visit, Day -3 prior to the single dose of enasidenib and at 0.5, 1, 2, 3, 4, 6, 8, and 10 hours post-dose.
Population: Participants who received 1 dose of enasidenib on Day -3 with sufficient data to determine PD parameters. Participants who received 2 doses on Day -3 or who received the incorrect dose were excluded. Participants in the Phase 1 Escalation BID and QD cohorts and Phase 1 Expansion cohorts were were grouped by dose for Day -3 analyses.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Enasidenib 30 mg | Enasidenib 50 mg | Enasidenib 75 mg | Enasidenib 100 mg | Enasidenib 150 mg | Enasidenib 200 mg | Enasidenib 300 mg | Enasidenib 450 mg | Enasidenib 650 mg
Number analyzed (Participants) | 3 | 7 | 7 | 56 | 8 | 10 | 4 | 1 | 1
percent change | 2.43 (1044.2) | -13.55 (71.3) | 9.32 (862.2) | -7.28 (270.8) | -16.61 (127.7) | -11.92 (95.3) | -17.79 (92.0) | -8.92 (NA) — Could not be calculated when N = 1 | -16.14 (NA) — Could not be calculated when N = 1

84. Secondary Outcome: Phase 1: Minimum Percent Change From Baseline Response Value Post-dose Over 10 Hours (%BRmin) for 2-HG After a Single Oral Dose of Enasidenib on Day -3
Description: The first 3 participants enrolled in each cohort of the dose escalation phase and the first 15 participants enrolled in each arm of Phase 1 Expansion received a single dose of enasidenib three days prior to starting the 28-day dosing regimen (Day -3). Plasma 2-HG was measured using qualified LC-MS/MS in order to characterize the pharmacodynamic (PD) effects of enasidenib; the LLOQ was 30.0 ng/mL. Minimum percent change from Baseline response value post-dose over 10 hours was calculated as: (minimum observed concentration post-dose over 10 hours [Rmin] - Baseline) / Baseline * 100. Baseline was equal to the average of the Screening and Day -3 (predose) 2-HG values. Data reported are the arithmetic mean and relative standard deviation expressed as a percentage.
Time Frame: Screening visit, Day -3 prior to the single dose of enasidenib and at 0.5, 1, 2, 3, 4, 6, 8, and 10 hours post-dose.
Population: Participants who received 1 dose of enasidenib on Day -3 with sufficient data to determine PD parameters. Participants who received 2 doses on Day -3 or who received the incorrect dose were excluded. Participants in the Phase 1 Dose Escalation BID and QD cohorts and Phase 1 Expansion cohorts were were grouped by dose for Day -3 analyses.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Enasidenib 30 mg | Enasidenib 50 mg | Enasidenib 75 mg | Enasidenib 100 mg | Enasidenib 150 mg | Enasidenib 200 mg | Enasidenib 300 mg | Enasidenib 450 mg | Enasidenib 650 mg
Number analyzed (Participants) | 4 | 9 | 9 | 57 | 8 | 11 | 4 | 2 | 1
percent change | -36.9 (43.9) | -37.7 (63.9) | -38.6 (96.4) | -47.5 (53.1) | -59.6 (44.5) | -56.9 (37.5) | -74.7 (9.0) | -31.5 (38.6) | -36.9 (NA) — Could not be calculated for N = 1

85. Secondary Outcome: Phase 1: Time of Minimum Observed Concentration Over 72 Hours Postdose (Tmin) of 2-HG After a Single Oral Dose of Enasidenib on Day -3
Description: The first 3 participants enrolled in each cohort of the dose escalation phase and the first 15 participants enrolled in each arm of Phase 1 Expansion received a single dose of enasidenib three days prior to starting the 28-day dosing regimen (Day -3). Plasma 2-HG was measured using qualified LC-MS/MS, the LLOQ was 30.0 ng/mL.
Time Frame: Day -3 prior to the single dose of enasidenib and at 0.5, 1, 2, 3, 4, 6, 8, 10, 24, 48, and 72 hours post-dose.
Population: as for outcome 83
Measure: Median (Full Range); unit: hours
Arm/Group | Enasidenib 30 mg | Enasidenib 50 mg | Enasidenib 75 mg | Enasidenib 100 mg | Enasidenib 150 mg | Enasidenib 200 mg | Enasidenib 300 mg | Enasidenib 450 mg | Enasidenib 650 mg
Number analyzed (Participants) | 4 | 9 | 9 | 57 | 8 | 11 | 4 | 2 | 1
hours | 35.78 [24.00 to 72.38] | 8.00 [1.13 to 72.42] | 23.92 [2.92 to 71.42] | 48.00 [0.50 to 73.58] | 48.20 [1.00 to 72.30] | 48.70 [6.07 to 72.45] | 48.10 [24.42 to 72.17] | 30.79 [13.33 to 48.25] | 8.17 [8.17 to 8.17]

86. Secondary Outcome: Phase 1: Percent Change From Baseline for Area Under the Effect Concentration Time Curve From Time 0 to 10 Hours Postdose of 2-HG After Multiple Oral Doses of Enasidenib
Description: Plasma 2-HG was measured using qualified LC-MS/MS, the LLOQ was 30.0 ng/mL. Area under the effect concentration time curve from time point zero (predose) up to 10 hours postdose (AUEC0-10) was calculated using the linear trapezoid rule. Percent change from baseline for AUEC0-10 was calculated as: (AUEC0-10 minus [Baseline*Tlast]) / (Baseline*Tlast) * 100, where Tlast corresponded to 10 hours and Baseline was equal to the average of the Screening and Day -3 (predose) 2-HG values. Data reported are the arithmetic mean and relative standard deviation expressed as a percentage.
Time Frame: Cycle 1, Day 15 and Cycle 2, Day 1 at predose and 0.5, 1, 2, 3, 4, 6, 8, and 10 hours post-dose.
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Enasidenib 30 mg BID | Enasidenib 50 mg BID | Enasidenib 75 mg BID | Enasidenib 100 mg BID | Enasidenib 150 mg BID | Enasidenib 50 mg QD | Phase 1 Dose Escalation: Enasidenib 75 mg QD | Phase 1 Dose Escalation: Enasidenib 100 mg QD | Phase 1 Dose Escalation: Enasidenib 150 mg QD | Phase 1 Dose Escalation: Enasidenib 200 mg QD | Phase 1 Dose Escalation: Enasidenib 300 mg QD | Phase 1 Dose Escalation: Enasidenib 450 mg QD | Phase 1 Dose Escalation: Enasidenib 650 mg QD
Number analyzed (Participants) | 6 | 7 | 6 | 5 | 4 | 5 | 6 | 89 | 5 | 10 | 7 | 4 | 2
percent change
  Cycle 1, Day 15: number analyzed (Participants) | 6 | 5 | 6 | 5 | 4 | 5 | 6 | 77 | 5 | 10 | 3 | 4 | 1
  Cycle 1, Day 15 | -62.18 (48.9) | -62.60 (113.1) | -87.19 (21.4) | -84.24 (14.2) | -79.40 (13.7) | -58.76 (44.9) | -69.00 (38.8) | -64.23 (80.3) | -71.67 (72.6) | -79.34 (34.1) | -87.74 (5.7) | -62.89 (48.8) | 2.54 (NA) — Could not be calculated for N = 1
  Cycle 2, Day 1: number analyzed (Participants) | 4 | 7 | 5 | 3 | 4 | 4 | 4 | 89 | 5 | 8 | 7 | 4 | 2
  Cycle 2, Day 1 | -49.01 (115.4) | -35.49 (430.9) | -64.63 (74.7) | -83.93 (19.0) | -78.07 (17.2) | -81.51 (25.9) | -66.41 (70.5) | -53.46 (190.7) | -37.70 (317.5) | -27.70 (599.5) | -87.88 (9.4) | -76.98 (40.2) | -82.28 (24.9)

87. Secondary Outcome: Phase 1: Minimum Percent Change From Baseline Response Value Post-dose Over 10 Hours (%BRmin) for 2-HG After Multiple Oral Doses of Enasidenib
Description: Plasma 2-HG was measured using qualified LC-MS/MS, the LLOQ was 30.0 ng/mL. Minimum percent change from Baseline response value post-dose over 10 hours was calculated as: (minimum observed concentration post-dose over 10 hours [Rmin] - Baseline) / Baseline * 100. Baseline was equal to the average of the Screening and Day -3 (predose) 2-HG values. Data reported are the arithmetic mean and relative standard deviation expressed as a percentage.
Time Frame: Cycle 1, Day 15 and Cycle 2, Day 1 at predose and 0.5, 1, 2, 3, 4, 6, 8, and 10 hours post-dose.
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Enasidenib 30 mg BID | Enasidenib 50 mg BID | Enasidenib 75 mg BID | Enasidenib 100 mg BID | Enasidenib 150 mg BID | Enasidenib 50 mg QD | Phase 1 Dose Escalation: Enasidenib 75 mg QD | Phase 1 Dose Escalation: Enasidenib 100 mg QD | Phase 1 Dose Escalation: Enasidenib 150 mg QD | Phase 1 Dose Escalation: Enasidenib 200 mg QD | Phase 1 Dose Escalation: Enasidenib 300 mg QD | Phase 1 Dose Escalation: Enasidenib 450 mg QD | Phase 1 Dose Escalation: Enasidenib 650 mg QD
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 4 | 5 | 7 | 102 | 6 | 12 | 7 | 5 | 3
percent change
  Cycle 1, Day 15: number analyzed (Participants) | 6 | 7 | 6 | 6 | 4 | 5 | 7 | 81 | 6 | 12 | 4 | 4 | 1
  Cycle 1, Day 15 | -69.0 (42.0) | -76.5 (56.4) | -89.2 (18.9) | -88.6 (12.3) | -81.4 (11.6) | -63.3 (40.7) | -79.3 (22.0) | -71.0 (57.1) | -80.4 (45.7) | -86.0 (25.3) | -91.2 (4.0) | -71.3 (31.5) | -23.1 (NA) — Could not be calculated for N = 1
  Cycle 2, Day 1: number analyzed (Participants) | 4 | 7 | 5 | 3 | 4 | 5 | 4 | 102 | 5 | 8 | 7 | 5 | 3
  Cycle 2, Day 1 | -54.8 (94.7) | -54.5 (192.9) | -68.9 (63.3) | -89.5 (12.5) | -80.7 (14.5) | -84.8 (18.5) | -70.6 (61.8) | -65.6 (94.7) | -47.2 (224.0) | -35.6 (422.0) | -89.8 (8.0) | -60.6 (83.8) | -53.5 (120.5)

88. Secondary Outcome: Phase 1: Time of Minimum Observed Concentration Over 10 Hours Postdose (Tmin) of 2-HG After Multiple Oral Doses of Enasidenib
Description: Plasma 2-HG was measured using qualified LC-MS/MS, the LLOQ was 30.0 ng/mL.
Time Frame: Cycle 1, Day 15 and Cycle 2, Day 1 at predose and 0.5, 1, 2, 3, 4, 6, 8, and 10 hours post-dose.
Population: Participants who received enasidenib on Cycle 1, Day 15 or Cycle 2, Day 1 with sufficient data to determine PD parameters. Participants who took less than 80% of their planned continuous dosing regimen were excluded from the analysis. Participants in the Phase 1 Escalation and Expansion Enasidenib 100 mg QD cohorts were combined for analysis.
Measure: Median (Full Range); unit: hours
Arm/Group | Enasidenib 30 mg BID | Enasidenib 50 mg BID | Enasidenib 75 mg BID | Enasidenib 100 mg BID | Enasidenib 150 mg BID | Enasidenib 50 mg QD | Phase 1 Dose Escalation: Enasidenib 75 mg QD | Phase 1 Dose Escalation: Enasidenib 100 mg QD | Phase 1 Dose Escalation: Enasidenib 150 mg QD | Phase 1 Dose Escalation: Enasidenib 200 mg QD | Phase 1 Dose Escalation: Enasidenib 300 mg QD | Phase 1 Dose Escalation: Enasidenib 450 mg QD | Phase 1 Dose Escalation: Enasidenib 650 mg QD
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 4 | 5 | 7 | 102 | 6 | 12 | 7 | 5 | 3
hours
  Cycle 1, Day 15: number analyzed (Participants) | 6 | 7 | 6 | 6 | 4 | 5 | 7 | 81 | 6 | 12 | 4 | 4 | 1
  Cycle 1, Day 15 | 4.00 [2.15 to 10.00] | 5.90 [1.00 to 10.00] | 3.03 [0.50 to 10.00] | 4.44 [1.10 to 10.00] | 1.00 [0.50 to 2.00] | 3.00 [0.50 to 6.05] | 5.85 [0.42 to 10.00] | 3.10 [0.35 to 10.00] | 6.50 [1.00 to 10.02] | 1.53 [0.50 to 8.00] | 7.08 [3.00 to 10.00] | 4.00 [0.50 to 8.07] | 2.87 [2.87 to 2.87]
  Cycle 2, Day 1: number analyzed (Participants) | 4 | 7 | 5 | 3 | 4 | 5 | 4 | 102 | 5 | 8 | 7 | 5 | 3
  Cycle 2, Day 1 | 0.98 [0.42 to 4.00] | 3.00 [1.00 to 10.00] | 6.17 [2.00 to 8.08] | 6.00 [0.97 to 6.00] | 2.00 [0.50 to 9.97] | 2.95 [0.48 to 10.08] | 6.96 [2.00 to 10.02] | 3.65 [0.30 to 10.32] | 4.00 [0.97 to 10.03] | 5.95 [1.00 to 7.93] | 7.92 [0.98 to 9.87] | 6.00 [1.00 to 9.83] | 2.00 [0.53 to 4.00]

ADVERSE EVENTS:
Time Frame: All cause Mortality, SAEs and Non SAEs were collected from first dose of IP to 28 days after last dose (Up to approximately 100 months)
Description: All cause Mortality, SAEs and Non SAEs was collected for treated population. A participant in Arm 2 was transferred to Arm 1 due to technical reasons after primary completion date and data collection for safety was conducted in the same arm.
Groups:
- Ph1Exp Arm 1 (R/R AML Age >=60 or R From BMT): Participants ≥ 60 years old with relapsed, refractory (R/R) AML or participants of any age if relapsed post-bone marrow transplant (BMT) received 100 mg enasidenib QD on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Ph1Exp Arm 2 (R/R AML Excluding Arm 1): Participants < 60 years old with R/R AML, excluding participants who relapsed post-BMT, received 100 mg enasidenib QD on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Ph1Exp Arm 3 (Untrt AML Age >=60 No SOC Chemo): Untreated AML participants ≥ 60 years old who declined standard of care received 100 mg enasidenib QD on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
- Ph1Exp Arm 4 (Not Eligible for Arms 1 to 3): Participants with advanced hematologic malignancies not eligible for Arms 1 to 3 received 100 mg enasidenib QD on Day 1 to Day 28 of each 28-day treatment cycle until disease progression or development of unacceptable toxicity.
Arm/Group | Phase 1 Dose Escalation: Enasidenib 30 mg BID | Phase 1 Dose Escalation: Enasidenib 50 mg BID | Phase 1 Dose Escalation: Enasidenib 75 mg BID | Phase 1 Dose Escalation: Enasidenib 100 mg BID | Phase 1 Dose Escalation: Enasidenib 150 mg BID | Phase 1 Dose Escalation: Enasidenib 50 mg QD | Phase 1 Dose Escalation: Enasidenib 75 mg QD | Phase 1 Dose Escalation: Enasidenib 100 mg QD | Phase 1 Dose Escalation: Enasidenib 150 mg QD | Phase 1 Dose Escalation: Enasidenib 200 mg QD | Phase 1 Dose Escalation: Enasidenib 300 mg QD | Phase 1 Dose Escalation: Enasidenib 450 mg QD | Phase 1 Dose Escalation: Enasidenib 650 mg QD | Ph1Exp Arm 1 (R/R AML Age >=60 or R From BMT) | Ph1Exp Arm 2 (R/R AML Excluding Arm 1) | Ph1Exp Arm 3 (Untrt AML Age >=60 No SOC Chemo) | Ph1Exp Arm 4 (Not Eligible for Arms 1 to 3) | Phase 2: Enasidenib 100 mg QD
All-Cause Mortality (participants affected / at risk) | 6/7 | 3/7 | 7/7 | 5/8 | 3/5 | 8/9 | 6/7 | 20/22 | 4/6 | 7/14 | 8/9 | 3/5 | 5/7 | 40/50 | 15/24 | 20/25 | 17/27 | 83/106
Serious Adverse Events (participants affected / at risk) | 6/7 | 6/7 | 6/7 | 7/8 | 3/5 | 9/9 | 5/7 | 19/22 | 4/6 | 11/14 | 7/9 | 5/5 | 6/7 | 43/50 | 18/24 | 20/25 | 20/27 | 86/106
Other Adverse Events (participants affected / at risk) | 7/7 | 7/7 | 7/7 | 8/8 | 5/5 | 8/9 | 7/7 | 22/22 | 6/6 | 14/14 | 9/9 | 5/5 | 7/7 | 50/50 | 23/24 | 25/25 | 27/27 | 106/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 Dose Escalation: Enasidenib 30 mg BID (N=7) | Phase 1 Dose Escalation: Enasidenib 50 mg BID (N=7) | Phase 1 Dose Escalation: Enasidenib 75 mg BID (N=7) | Phase 1 Dose Escalation: Enasidenib 100 mg BID (N=8) | Phase 1 Dose Escalation: Enasidenib 150 mg BID (N=5) | Phase 1 Dose Escalation: Enasidenib 50 mg QD (N=9) | Phase 1 Dose Escalation: Enasidenib 75 mg QD (N=7) | Phase 1 Dose Escalation: Enasidenib 100 mg QD (N=22) | Phase 1 Dose Escalation: Enasidenib 150 mg QD (N=6) | Phase 1 Dose Escalation: Enasidenib 200 mg QD (N=14) | Phase 1 Dose Escalation: Enasidenib 300 mg QD (N=9) | Phase 1 Dose Escalation: Enasidenib 450 mg QD (N=5) | Phase 1 Dose Escalation: Enasidenib 650 mg QD (N=7) | Ph1Exp Arm 1 (R/R AML Age >=60 or R From BMT) (N=50) | Ph1Exp Arm 2 (R/R AML Excluding Arm 1) (N=24) | Ph1Exp Arm 3 (Untrt AML Age >=60 No SOC Chemo) (N=25) | Ph1Exp Arm 4 (Not Eligible for Arms 1 to 3) (N=27) | Phase 2: Enasidenib 100 mg QD (N=106)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 2 | 5
BONE MARROW FAILURE (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
FEBRILE BONE MARROW APLASIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 4 | 1 | 1 | 1 | 6 | 0 | 9 | 2 | 1 | 2 | 1 | 0 | 16 | 5 | 3 | 3 | 35
HAEMOLYSIS (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 3 | 1 | 3 | 0 | 0 | 2 | 4 | 1 | 1 | 0 | 13
LEUKOSTASIS SYNDROME (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
LYMPHADENITIS (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
SPLEEN DISORDER (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
SPLENIC INFARCTION (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
SPLENIC VEIN THROMBOSIS (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 4
THROMBOCYTOSIS (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
ANGINA PECTORIS (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 1 | 1
ATRIAL FLUTTER (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ATRIOVENTRICULAR BLOCK FIRST DEGREE (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
CARDIAC ARREST (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
CARDIAC FAILURE (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
CARDIAC TAMPONADE (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
CARDIAC VALVE DISEASE (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
CARDIOPULMONARY FAILURE (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
DIASTOLIC DYSFUNCTION (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
PERICARDIAL EFFUSION (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
PERICARDITIS (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
APLASIA (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ARTERIOVENOUS MALFORMATION (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
RETINAL HAEMORRHAGE (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
APPENDIX DISORDER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
COLITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
CONSTIPATION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 1 | 1 | 6
DUODENAL ULCER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
DYSPHAGIA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
ENTEROCOLITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
ENTEROVESICAL FISTULA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
GASTRIC ULCER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
GASTRITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 3 | 0 | 2
GASTROINTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
GINGIVAL BLEEDING (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ILEUS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
INTESTINAL PERFORATION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
INTRA-ABDOMINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MELAENA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
MOUTH ULCERATION (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 2 | 0 | 2 | 5
NEUTROPENIC COLITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OEDEMA MOUTH (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OESOPHAGITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
PERIODONTAL DISEASE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
PROCTALGIA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
SMALL INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
STOMATITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 1 | 2
VOMITING (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 1 | 4
ASTHENIA (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
CATHETER SITE HAEMORRHAGE (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
CHEST PAIN (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CHILLS (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
FACIAL PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
FATIGUE (General disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 8
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
HYPOTHERMIA (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
LOCALISED OEDEMA (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MALAISE (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
MASS (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
MUCOSAL INFLAMMATION (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 6
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
OEDEMA PERIPHERAL (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
PYREXIA (General disorders) | 0 | 2 | 2 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 1 | 0 | 4 | 1 | 2 | 2 | 11
SECRETION DISCHARGE (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
SUDDEN DEATH (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ACUTE HEPATIC FAILURE (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HEPATIC CYTOLYSIS (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HEPATIC STEATOSIS (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
HYPERTRANSAMINASAEMIA (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
GRAFT VERSUS HOST DISEASE (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
HAEMOPHAGOCYTIC LYMPHOHISTIOCYTOSIS (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
ABDOMINAL ABSCESS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
ABSCESS BACTERIAL (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ABSCESS LIMB (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ANORECTAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
APPENDICITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
ARTHRITIS BACTERIAL (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
ASPERGILLUS INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BACTERAEMIA (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 4
BACTERIAL SEPSIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
CELLULITIS (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 1 | 3
CLOSTRIDIAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 1 | 0 | 5
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 0
CYSTITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
DEVICE RELATED INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 1
DIARRHOEA INFECTIOUS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
DIVERTICULITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
ENCEPHALITIS VIRAL (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ENTEROCOCCAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
ENTEROCOCCAL SEPSIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
GASTROENTERITIS VIRAL (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
GINGIVITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
GRANULICATELLA INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
GROIN ABSCESS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
INFLUENZA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
KLEBSIELLA SEPSIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
LARGE INTESTINE INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
LOCALISED INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
LUNG ABSCESS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
LYMPH GLAND INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
MICROCOCCUS INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OESOPHAGEAL CANDIDIASIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ORAL CANDIDIASIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OSTEOMYELITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
PERITONITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
PHARYNGITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
PNEUMONIA (Infections and infestations) | 2 | 2 | 1 | 2 | 1 | 3 | 0 | 3 | 0 | 4 | 1 | 1 | 1 | 13 | 10 | 6 | 6 | 26
PNEUMONIA ASPIRATION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
PNEUMONIA FUNGAL (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
PSOAS ABSCESS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PYELONEPHRITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
SCROTAL ABSCESS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
SCROTAL CELLULITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
SEPSIS (Infections and infestations) | 3 | 1 | 0 | 3 | 0 | 4 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 8 | 4 | 1 | 2 | 13
SEPTIC SHOCK (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
SINUSITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 4
SINUSITIS BACTERIAL (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
SINUSITIS FUNGAL (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
SKIN INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
STAPHYLOCOCCAL SKIN INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
URETHRAL ABSCESS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 3 | 0 | 1 | 5
URINARY TRACT INFECTION BACTERIAL (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
UROSEPSIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
VIRAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
VIRAL MYOCARDITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
FALL (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0
HEAD INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 6
WOUND HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
BLOOD BILIRUBIN INCREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1
BLOOD CREATINE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
BLOOD CULTURE POSITIVE (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
BLOOD LACTIC ACID INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
BLOOD PRESSURE SYSTOLIC DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
LIPASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
MENSTRUATION NORMAL (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OCCULT BLOOD POSITIVE (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PLATELET COUNT DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
PROTHROMBIN TIME PROLONGED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
TROPONIN I INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
TROPONIN INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
ACIDOSIS (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
HYPERVOLAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
IRON OVERLOAD (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 1 | 1 | 3 | 2 | 7
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 1
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MYOSITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
RHEUMATIC DISORDER (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
ANAL SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CHLOROMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DIFFERENTIATION SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 4 | 0 | 2 | 1 | 1 | 1 | 2 | 2 | 3 | 0 | 7
HAEMANGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
LYMPHOPROLIFERATIVE DISORDER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
CEREBRAL ISCHAEMIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
DIZZINESS (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
FACIAL PARALYSIS (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 1
HEADACHE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
INTRACRANIAL HAEMATOMA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
ISCHAEMIC STROKE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
NERVE COMPRESSION (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
PRESYNCOPE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
SCIATICA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
SEIZURE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
SYNCOPE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
ANXIETY (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 4
DEPRESSION (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
HALLUCINATION (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MANIA (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 4 | 2 | 3 | 1 | 5
AZOTAEMIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HAEMATURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
HYDRONEPHROSIS (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
PRERENAL FAILURE (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
RENAL FAILURE (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
SUBCAPSULAR RENAL HAEMATOMA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
PENILE PAIN (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
PROSTATITIS (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
SCROTAL OEDEMA (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 2 | 8
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
NASAL NECROSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
PHARYNGEAL INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 4
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 2 | 0 | 8
NEUTROPHILIC DERMATOSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
PYODERMA GANGRENOSUM (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
SKIN DISORDER (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HAEMORRHAGE PROPHYLAXIS (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
INCISIONAL DRAINAGE (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
EMBOLISM (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HAEMATOMA (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
HYPERTENSION (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
HYPOTENSION (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 2 | 6
HYPOVOLAEMIC SHOCK (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
LYMPHOEDEMA (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
SHOCK HAEMORRHAGIC (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 Dose Escalation: Enasidenib 30 mg BID (N=7) | Phase 1 Dose Escalation: Enasidenib 50 mg BID (N=7) | Phase 1 Dose Escalation: Enasidenib 75 mg BID (N=7) | Phase 1 Dose Escalation: Enasidenib 100 mg BID (N=8) | Phase 1 Dose Escalation: Enasidenib 150 mg BID (N=5) | Phase 1 Dose Escalation: Enasidenib 50 mg QD (N=9) | Phase 1 Dose Escalation: Enasidenib 75 mg QD (N=7) | Phase 1 Dose Escalation: Enasidenib 100 mg QD (N=22) | Phase 1 Dose Escalation: Enasidenib 150 mg QD (N=6) | Phase 1 Dose Escalation: Enasidenib 200 mg QD (N=14) | Phase 1 Dose Escalation: Enasidenib 300 mg QD (N=9) | Phase 1 Dose Escalation: Enasidenib 450 mg QD (N=5) | Phase 1 Dose Escalation: Enasidenib 650 mg QD (N=7) | Ph1Exp Arm 1 (R/R AML Age >=60 or R From BMT) (N=50) | Ph1Exp Arm 2 (R/R AML Excluding Arm 1) (N=24) | Ph1Exp Arm 3 (Untrt AML Age >=60 No SOC Chemo) (N=25) | Ph1Exp Arm 4 (Not Eligible for Arms 1 to 3) (N=27) | Phase 2: Enasidenib 100 mg QD (N=106)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 4 | 2 | 1 | 2 | 2 | 2 | 6 | 1 | 4 | 2 | 2 | 2 | 11 | 4 | 11 | 6 | 40
BLOOD LOSS ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COAGULOPATHY (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 2
EOSINOPHILIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 5 | 1 | 2 | 2 | 0 | 0 | 2 | 3 | 1 | 1 | 9
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 5 | 1 | 2 | 1 | 0 | 0 | 6 | 6 | 2 | 0 | 15
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 3 | 1 | 3
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 1
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 2 | 1 | 2 | 1 | 4 | 2 | 1 | 0 | 10
SPLENOMEGALY (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 3 | 1 | 2 | 1 | 1 | 2 | 1 | 4 | 1 | 3 | 2 | 1 | 2 | 7 | 5 | 4 | 7 | 25
THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
THROMBOCYTOSIS (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ACUTE LEFT VENTRICULAR FAILURE (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 4
BUNDLE BRANCH BLOCK RIGHT (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CARDIAC FAILURE (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
CARDIAC VALVE DISEASE (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DIASTOLIC DYSFUNCTION (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PALPITATIONS (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 4
PERICARDIAL EFFUSION (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 3
SINUS BRADYCARDIA (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3
SINUS TACHYCARDIA (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 2
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
SYSTOLIC DYSFUNCTION (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TACHYCARDIA (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 0 | 1 | 5
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
APLASIA (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
GILBERT'S SYNDROME (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
HYDROCELE (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
DEAFNESS (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1
EAR CONGESTION (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
EAR DISCOMFORT (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
EAR DISORDER (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
EAR PAIN (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
EXCESSIVE CERUMEN PRODUCTION (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HYPOACUSIS (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
TINNITUS (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
VERTIGO (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
ADRENAL HAEMATOMA (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ADRENAL MASS (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
CATARACT (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
CHALAZION (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1
CONJUNCTIVAL HYPERAEMIA (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DIPLOPIA (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
DRY EYE (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 4
EYE DISCHARGE (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
EYE IRRITATION (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
EYE PAIN (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
EYE SWELLING (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
LACRIMATION INCREASED (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3
OCULAR HYPERAEMIA (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ORBITAL HAEMATOMA (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
VISION BLURRED (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 6
VISUAL ACUITY REDUCED (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 1 | 3 | 1 | 0 | 3 | 2 | 3 | 0 | 3 | 1 | 1 | 1 | 5 | 4 | 5 | 2 | 13
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 4 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 8
ANAL INCONTINENCE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ANOGENITAL DYSPLASIA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
APHTHOUS ULCER (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
CHRONIC GASTRITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
COLITIS (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 4
CONSTIPATION (Gastrointestinal disorders) | 1 | 2 | 2 | 2 | 2 | 6 | 2 | 4 | 2 | 4 | 2 | 0 | 3 | 16 | 7 | 10 | 5 | 27
DIARRHOEA (Gastrointestinal disorders) | 2 | 3 | 3 | 4 | 2 | 5 | 3 | 10 | 3 | 7 | 3 | 4 | 4 | 20 | 6 | 7 | 11 | 42
DRY MOUTH (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 8
DUODENOGASTRIC REFLUX (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DYSPEPSIA (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 4 | 0 | 0 | 1 | 1 | 2 | 5 | 3 | 2 | 2 | 5
DYSPHAGIA (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 5 | 0 | 2 | 1 | 1
ENTEROCOLITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
FAECES DISCOLOURED (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
FLATULENCE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 5
FREQUENT BOWEL MOVEMENTS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
GASTRITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 2
GASTROINTESTINAL ANGIECTASIA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 4 | 2 | 1 | 0 | 0 | 0 | 3 | 2 | 1 | 2 | 5
GINGIVAL BLEEDING (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 1 | 0 | 1 | 3 | 4 | 2 | 2 | 6
GINGIVAL HYPERTROPHY (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 4 | 2 | 0 | 0 | 0
GINGIVAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
GLOSSITIS (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 3 | 0 | 1 | 0 | 0 | 1 | 4 | 1 | 0 | 1 | 7
ILEUS (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
INTRA-ABDOMINAL HAEMATOMA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
LIP DISORDER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
MOUTH HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1
MOUTH ULCERATION (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
NAUSEA (Gastrointestinal disorders) | 3 | 5 | 2 | 4 | 2 | 5 | 4 | 7 | 3 | 9 | 4 | 2 | 2 | 21 | 13 | 9 | 12 | 58
ODYNOPHAGIA (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
OESOPHAGITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
ORAL BLOOD BLISTER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
ORAL DISORDER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 2
ORAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 2
POOR DENTAL CONDITION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PROCTALGIA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
RETCHING (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
SALIVARY HYPERSECRETION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
STOMATITIS (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 8
TONGUE COATED (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TOOTHACHE (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 3
VOMITING (Gastrointestinal disorders) | 2 | 4 | 1 | 3 | 2 | 2 | 4 | 3 | 4 | 6 | 3 | 1 | 2 | 20 | 8 | 7 | 4 | 33
ASTHENIA (General disorders) | 0 | 5 | 2 | 1 | 1 | 1 | 3 | 5 | 1 | 3 | 0 | 1 | 0 | 10 | 2 | 2 | 2 | 14
AXILLARY PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
CATHETER SITE EROSION (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CATHETER SITE HAEMORRHAGE (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
CATHETER SITE IRRITATION (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CATHETER SITE PAIN (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CHEST DISCOMFORT (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
CHEST PAIN (General disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 2 | 2 | 3 | 5
CHILLS (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 2 | 3 | 7
CYST (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
FACE OEDEMA (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
FATIGUE (General disorders) | 2 | 1 | 2 | 3 | 3 | 3 | 3 | 7 | 1 | 6 | 3 | 3 | 4 | 18 | 12 | 12 | 10 | 48
GAIT DISTURBANCE (General disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HERNIA (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
IMPAIRED HEALING (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
INFUSION SITE ERYTHEMA (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
INFUSION SITE INDURATION (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
LOCALISED OEDEMA (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
MALAISE (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 2 | 1
MASS (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
MUCOSAL DISCOLOURATION (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MUCOSAL INFLAMMATION (General disorders) | 2 | 1 | 4 | 1 | 1 | 0 | 0 | 5 | 0 | 1 | 0 | 1 | 0 | 7 | 4 | 2 | 0 | 10
NODULE (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
OEDEMA (General disorders) | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 10
OEDEMA PERIPHERAL (General disorders) | 3 | 2 | 3 | 4 | 1 | 2 | 1 | 3 | 3 | 5 | 1 | 1 | 2 | 17 | 3 | 11 | 5 | 34
PAIN (General disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 4 | 2 | 0 | 1 | 8
PERIPHERAL SWELLING (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
PRE-EXISTING CONDITION IMPROVED (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PYREXIA (General disorders) | 2 | 5 | 1 | 1 | 0 | 2 | 2 | 7 | 2 | 6 | 1 | 2 | 2 | 12 | 6 | 2 | 6 | 25
SWELLING (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0
SWELLING FACE (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
TEMPERATURE INTOLERANCE (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
XEROSIS (General disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
CHOLESTASIS (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 2
HEPATIC CYTOLYSIS (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
HEPATOMEGALY (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
HEPATOSPLENOMEGALY (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 6 | 1 | 3 | 3 | 9
JAUNDICE (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
OCULAR ICTERUS (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
GRAFT VERSUS HOST DISEASE (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
SEASONAL ALLERGY (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ANAL ABSCESS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BACTERAEMIA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2
BACTERIAL COLITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BONE ABSCESS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BRONCHITIS (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
CANDIDA INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 2
CATHETER SITE INFECTION (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
CELLULITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 3 | 0 | 2 | 3
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 4
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 2
CONJUNCTIVITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 2
CONJUNCTIVITIS BACTERIAL (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
DEVICE RELATED INFECTION (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
EAR INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
FOLLICULITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
FUNGAL INFECTION (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
FURUNCLE (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
GASTROINTESTINAL FUNGAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
GASTROINTESTINAL VIRAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
GENITAL HERPES (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
GENITAL INFECTION FUNGAL (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
GINGIVITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0
HAEMORRHOID INFECTION (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
INCISION SITE CELLULITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
INFECTION (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
INFLUENZA (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 4
KLEBSIELLA BACTERAEMIA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
LUNG ABSCESS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MUCOSAL INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
NAIL BED INFECTION BACTERIAL (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
NASOPHARYNGITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1
OESOPHAGEAL CANDIDIASIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ORAL CANDIDIASIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 4
ORAL HERPES (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
PARONYCHIA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
PHARYNGITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
PNEUMONIA (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 2 | 2 | 2 | 0 | 2 | 0 | 1 | 0 | 7 | 4 | 3 | 1 | 15
PNEUMONIA FUNGAL (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2
PSEUDOMONAS INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PULPITIS DENTAL (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
RASH PUSTULAR (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
RHINITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
SEPSIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 5
SINUSITIS (Infections and infestations) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 5
SINUSITIS FUNGAL (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
SKIN INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 3 | 2
STENOTROPHOMONAS INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TOOTH ABSCESS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
TOOTH INFECTION (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 6 | 0 | 3 | 4 | 5
URINARY TRACT INFECTION (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 7 | 1 | 2 | 2 | 5
URINARY TRACT INFECTION FUNGAL (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
VAGINAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
VIRAL RHINITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
WOUND INFECTION STAPHYLOCOCCAL (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ANIMAL SCRATCH (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
CONTUSION (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 3 | 1 | 1 | 0 | 0 | 2 | 2 | 0 | 1 | 3 | 8
EYE CONTUSION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 2 | 3 | 1 | 3 | 1 | 2 | 1 | 1 | 1 | 7 | 1 | 5 | 2 | 11
HEAD INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
JOINT INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PERIORBITAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
POST PROCEDURAL DISCHARGE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
POST-TRAUMATIC PAIN (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 2
REACTIVE GASTROPATHY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
STRESS FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TOOTH FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3
WOUND (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 4
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 1 | 2 | 5 | 3 | 3 | 3 | 13
AMYLASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 3 | 0 | 1 | 3 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 6 | 1 | 4 | 5 | 15
BILIRUBIN CONJUGATED INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 1 | 2 | 1 | 4 | 1 | 3 | 1 | 2
BLOOD BILIRUBIN INCREASED (Investigations) | 1 | 3 | 2 | 3 | 3 | 1 | 3 | 9 | 4 | 8 | 2 | 4 | 4 | 20 | 8 | 8 | 8 | 23
BLOOD BILIRUBIN UNCONJUGATED INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
BLOOD CREATINE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
BLOOD CREATININE INCREASED (Investigations) | 0 | 0 | 2 | 1 | 0 | 2 | 0 | 2 | 2 | 0 | 1 | 0 | 2 | 6 | 2 | 5 | 4 | 13
BLOOD FIBRINOGEN DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 3
BLOOD PHOSPHORUS INCREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 1
BLOOD PRESSURE DECREASED (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BLOOD UREA INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 2
BLOOD URIC ACID INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
BRAIN NATRIURETIC PEPTIDE INCREASED (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CARBON DIOXIDE DECREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
EJECTION FRACTION DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 2 | 0 | 0 | 0 | 3 | 3 | 3 | 0 | 4
EPSTEIN-BARR VIRUS ANTIBODY POSITIVE (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
HAEMOGLOBIN DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
HEPATIC ENZYME INCREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HUMAN METAPNEUMOVIRUS TEST POSITIVE (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
IMMUNOGLOBULINS DECREASED (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
LIPASE INCREASED (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 1 | 3 | 0 | 1 | 1 | 3 | 3 | 0
LYMPHOCYTE COUNT DECREASED (Investigations) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 6
LYMPHOCYTE COUNT INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
MAMMOGRAM ABNORMAL (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MYOCARDIAL NECROSIS MARKER INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
NEUTROPHIL COUNT DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 4 | 1 | 3
NEUTROPHIL COUNT INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
OXYGEN SATURATION DECREASED (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
PLATELET COUNT DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 6 | 2 | 5 | 2 | 11
PLATELET COUNT INCREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
PROTEIN TOTAL INCREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PROTHROMBIN LEVEL DECREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PROTHROMBIN TIME PROLONGED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
URINE OUTPUT DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
WEIGHT DECREASED (Investigations) | 0 | 0 | 1 | 2 | 3 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 12 | 2 | 2 | 3 | 12
WEIGHT INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 2
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 2 | 3 | 1 | 5
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 2 | 1
CELL DEATH (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 3 | 2 | 3 | 3 | 2 | 3 | 1 | 9 | 2 | 5 | 1 | 4 | 1 | 24 | 9 | 10 | 9 | 22
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 6 | 1 | 3 | 0 | 6
GOUT (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 2 | 2 | 0 | 4 | 2 | 3 | 0 | 2 | 13
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 2 | 5
HYPERLIPASAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
HYPERMAGNESAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 1
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 | 3 | 1 | 1 | 2 | 1 | 0 | 5 | 0 | 1 | 2 | 0 | 1 | 5 | 2 | 1 | 2 | 8
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 3 | 2 | 1 | 0 | 2 | 3 | 1 | 1 | 3 | 0 | 1 | 12 | 6 | 4 | 8 | 15
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 1 | 0 | 2 | 2 | 2 | 3 | 2 | 7
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 | 2 | 1 | 3 | 1 | 1 | 2 | 5 | 1 | 2 | 2 | 2 | 4 | 9 | 5 | 5 | 2 | 17
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 3 | 2 | 1 | 1 | 3 | 2 | 6 | 1 | 3 | 4 | 1 | 2 | 13 | 9 | 8 | 7 | 28
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 | 3 | 2 | 1 | 0 | 2 | 0 | 3 | 1 | 3 | 2 | 1 | 2 | 8 | 4 | 6 | 7 | 20
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 2 | 2 | 3 | 6 | 4 | 5 | 3 | 8
HYPOPHAGIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 | 2 | 3 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 2 | 1 | 3 | 4 | 1 | 12
HYPOPROTEINAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
MALNUTRITION (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
STEROID DIABETES (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 4 | 2 | 2 | 1 | 5 | 0 | 3 | 2 | 2 | 0 | 8 | 4 | 1 | 7 | 23
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 4 | 0 | 1 | 1 | 3 | 1 | 1 | 2 | 3 | 1 | 6 | 3 | 4 | 4 | 18
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 3 | 3 | 0 | 1 | 6
CERVICAL SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
CHONDROCALCINOSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CHONDROPATHY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
JOINT RANGE OF MOTION DECREASED (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 1 | 1
MOBILITY DECREASED (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 3 | 1 | 3 | 1 | 5
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 3 | 1 | 12
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 6 | 0 | 1 | 0 | 0 | 0 | 6 | 2 | 0 | 4 | 5
MYOSITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 2 | 3 | 0 | 1 | 3
OSTEITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OSTEOPENIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 4 | 1 | 2 | 1 | 1 | 0 | 4 | 0 | 1 | 0 | 1 | 1 | 4 | 2 | 3 | 3 | 15
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
SPINAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TENDON PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TENDONITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
BOWEN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DIFFERENTIATION SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 0 | 8
HAEMANGIOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MELANOCYTIC NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
VULVAL CANCER STAGE 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
AGEUSIA (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
APHASIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
DIZZINESS (Nervous system disorders) | 1 | 1 | 0 | 2 | 0 | 3 | 0 | 5 | 0 | 1 | 0 | 2 | 1 | 9 | 2 | 7 | 2 | 14
DYSGEUSIA (Nervous system disorders) | 0 | 0 | 1 | 2 | 2 | 0 | 1 | 3 | 1 | 1 | 0 | 1 | 0 | 7 | 2 | 2 | 3 | 11
HEADACHE (Nervous system disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 6 | 1 | 4 | 1 | 1 | 1 | 9 | 6 | 4 | 5 | 27
HEMIPARESIS (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HYPERAESTHESIA (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HYPOAESTHESIA (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1
LETHARGY (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
NERVOUS SYSTEM DISORDER (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
NEURALGIA (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 3 | 0 | 2 | 2 | 4
PARAESTHESIA (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 5 | 0 | 0 | 2 | 3
PAROSMIA (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 11
SCIATICA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SEIZURE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
SINUS HEADACHE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
SOMNOLENCE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SYNCOPE (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0
TASTE DISORDER (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
TOXIC ENCEPHALOPATHY (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
TREMOR (Nervous system disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2
ADJUSTMENT DISORDER (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ADJUSTMENT DISORDER WITH DEPRESSED MOOD (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
AGITATION (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2
ANGER (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ANXIETY (Psychiatric disorders) | 1 | 2 | 2 | 1 | 1 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 4 | 4 | 4 | 3 | 15
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 11
DELIRIUM (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 1 | 0 | 1 | 1
DEPRESSION (Psychiatric disorders) | 0 | 1 | 1 | 3 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 8 | 2 | 2 | 4 | 9
HALLUCINATION (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 3
HALLUCINATION, VISUAL (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
INSOMNIA (Psychiatric disorders) | 1 | 3 | 0 | 2 | 2 | 1 | 2 | 3 | 1 | 2 | 0 | 2 | 0 | 6 | 5 | 3 | 4 | 20
IRRITABILITY (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
LIBIDO DECREASED (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 1 | 0
MOOD SWINGS (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PSYCHOMOTOR RETARDATION (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SLEEP DISORDER (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TOBACCO WITHDRAWAL SYMPTOMS (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 2 | 1 | 2 | 2 | 10
BLADDER SPASM (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
CHROMATURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
DYSURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 3
HAEMATURIA (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
NOCTURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
POLLAKIURIA (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 5
POLYURIA (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
PROTEINURIA (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 3 | 0
RENAL FAILURE (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 2 | 0 | 5
RENAL TUBULAR DYSFUNCTION (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
URETEROLITHIASIS (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
URETHRITIS NONINFECTIVE (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
URINARY INCONTINENCE (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 6
URINARY RETENTION (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
BREAST PAIN (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
GENITAL LESION (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SCROTAL OEDEMA (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
SCROTAL PAIN (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TESTICULAR PAIN (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
VULVAL DISORDER (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 2 | 2 | 1 | 4 | 0 | 8 | 4 | 5 | 2 | 1 | 2 | 16 | 4 | 4 | 13 | 35
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2 | 2 | 2 | 5 | 3 | 8 | 2 | 0 | 3 | 1 | 2 | 15 | 3 | 10 | 10 | 37
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 1 | 3 | 1 | 3 | 1 | 3 | 0 | 0 | 3 | 6 | 2 | 5 | 1 | 21
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 3 | 6
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 6
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 3
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 3 | 1 | 3 | 0 | 2 | 2 | 0 | 0 | 6 | 1 | 2 | 4 | 9
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 2 | 2 | 5
OROPHARYNGEAL PLAQUE (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PARANASAL SINUS HYPERSECRETION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 2 | 2 | 1 | 1 | 4 | 2 | 3 | 0 | 6
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1
PULMONARY GRANULOMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 2
RALES (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
RESPIRATORY DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 1
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 2 | 4 | 2 | 3 | 1 | 4
RHONCHI (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2
SINUS PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TACHYPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
UPPER-AIRWAY COUGH SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 1
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 2
BLOOD BLISTER (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CAPILLARITIS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COLD SWEAT (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DERMAL CYST (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 3
DERMATITIS EXFOLIATIVE GENERALISED (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 5
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 5
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 0 | 0 | 2 | 7
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
HYPERTRICHOSIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
NAIL RIDGING (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 4
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
PAPULE (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
PETECHIAE (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 2 | 0 | 1 | 1 | 4 | 1 | 0 | 7
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 3 | 1 | 4 | 2 | 0 | 0 | 4 | 4 | 3 | 4 | 10
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
PURPURA (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
RASH (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 1 | 0 | 1 | 1 | 2 | 1 | 2 | 0 | 2 | 1 | 10 | 2 | 2 | 9 | 11
RASH MACULAR (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 2 | 0 | 0 | 4 | 0 | 3 | 4 | 15
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
RASH VESICULAR (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
SEBORRHOEIC DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SKIN DISCOLOURATION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
SKIN DISORDER (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SKIN INDURATION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SKIN IRRITATION (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SKIN LESION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 1 | 0 | 0 | 4 | 0 | 1 | 3 | 1
SKIN MASS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
SOLAR LENTIGO (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TOXIC SKIN ERUPTION (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
TOOTH EXTRACTION (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 2
EMBOLISM (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
HAEMATOMA (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 3 | 0 | 0 | 1 | 2
HAEMORRHAGE (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HOT FLUSH (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
HYPERTENSION (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 11
HYPOTENSION (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 3 | 0 | 1 | 1 | 1 | 1 | 13 | 3 | 1 | 0 | 12
LYMPHOCELE (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 1
PALLOR (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
SCALP HAEMATOMA (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
THROMBOPHLEBITIS (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
VARICOSE VEIN (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
1 participant was randomized in Arm 2 before Primary analysis in error. After primary completion , the decision was made to randomize the participant into Arm 1 from Arm 2. Only adverse events section is revised as per this randomization change.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication

DOCUMENTS (2):
  • Study Protocol (2017-10-17): https://cdn.clinicaltrials.gov/large-docs/98/NCT01915498/Prot_001.pdf
  • Statistical Analysis Plan (2019-10-04): https://cdn.clinicaltrials.gov/large-docs/98/NCT01915498/SAP_000.pdf